

# APL-B-021-13 (NCT03070964)

A Phase II Study of Plitidepsin in Patients with Relapsed or Refractory Angioimmunoblastic T-cell Lymphoma

STATISTICAL ANALYSIS PLAN

Version: 1.0

Date: 13-October-2016

# **TABLE OF CONTENTS**

| 1 | ST | UDY RATIONALE | 6 |
|---|---|---|---|
| 2 | ST | UDY DESIGN | |
| 3 | OB | JECTIVES AND ENDPOINTS | 7<br>8 |
| | 3.1 | Primary objective | |
| | 3.2 | Secondary objectives | 8 |
| | 3.3 | Endpoints | 8 |
| 4 | PA | TIENTS EVALUABILITY CRITERIA | 9 |
| | 4.1 | Analysis sets definitions | 9 |
| | | Efficacy populations | 10 |
| | 4.3 | J 1 1 | 10 |
| 5 | | MPLE CONSIDERATIONS | 10 |
| 6 | | ATISTICAL METHODOLOGY FOR EFFICACY | 11 |
| | 6.1 | Planned analyses and definitions | 11 |
| | 6.1 | J 1 J | 11 |
| | 6.1 | J 1 J | 11 |
| | 6.2 | Efficacy analysis methods | 12 |
| | | 1 Primary endpoint | 12 |
| | | 2 Secondary analyses | 12 |
| 7 | | ATISTICAL METHODOLOGY FOR SAFETY | 13 |
| | 7.1 | Toxicity and adverse events | 13 |
| | 7.2 | Clinical laboratory evaluation | 14 |
| | | Vital signs, physical examination, left ventricular ejection fraction (LVEF) and | |
| | | ocardiogram findings | 14 |
| _ | 7.4 | Deaths and other Serious Adverse Events | 14 |
| 8 | | HER ANALYSES | 14 |
| | 8.1 | Baseline and demographic data | 14 |
| | 8.2 | Treatment administration | 15 |
| | 8.3 | Subsequent therapy | 15 |
| | 8.4 | Protocol deviations | 15 |
| | 8.5 | Pharmacokinetic and biomarkers analyses | 15 |
| | 8.6 | Imputation of incomplete dates | 16 |
| | 8.7 | Subgroup analyses | 16 |
| | | Decimal places and methods for handling missing data | 17 |
| | 8.9 | Interim and group sequential analyses | 17 |
| ^ | 8.10 | Identification of fixed or random effects models | 17 |
| 9 | | ATISTICAL SOFTWARE | 17 |
| 1 / | | NDIX I | 18 |
| 1( | | dy Patients | 18 |
| | 10.1 | Patient disposition | 18 |
| | 10.2 | Reasons for treatment discontinuation | 19 |
| 1 - | 10.3 | Protocol deviations | 20 |
| 1. | | icacy Evaluation | 21 |
| | 11.1 | Demographic and other baseline characteristics | 21 |

| | 11.1.1 | Patient characteristics at baseline | 21 |
|---|---|---|---|
| | 11.1.2 | Local histopathological diagnosis | 21 |
| | 11.1.3 | Disease at diagnosis, time from diagnosis and current disease | 22 |
| | | Prior anticancer therapy | 24 |
| | 11.1.5 | ± 7 | 25 |
| | 11.1.6 | Physical examination, vital signs, electrocardiogram and other tests | 25 |
| | 11.1.7 | Hematological values at baseline | 28 |
| | 11.1.8 | • | 29 |
| | 11.1.9 | Other metabolic values at baseline | 29 |
| | 11.1.10 | | 30 |
| | 11.1.11 | | 30 |
| 1 | 1.2 | Measurements of treatment compliance | 31 |
| 1 | 1.3 | Efficacy analysis | 31 |
| | 11.3.1 | | 31 |
| | 11.3.2 | Secondary analyses | 32 |
| | 11.3.3 | Follow-up | 38 |
| | | Multivariate analyses | 39 |
| | | Best reduction in sum of the product of the diameters lesions | 42 |
| | 11.3.6 | Characteristics of responders | 42 |
| 12 | Safety A | • | 43 |
| 1. | 2.1 | Extent of exposure | 43 |
| | 12.1.1 | Treatment administration | 43 |
| | 12.1.2 | Cycle delays | 43 |
| | 12.1.3 | Dose omissions | 44 |
| | 12.1.4 | Dose reductions | 45 |
| | 12.1.5 | Infusions temporarily interrupted | 46 |
| | 12.1.6 | Prophylactic medication administration | 46 |
| 1. | 2.2 | Adverse Events (AEs) | 47 |
| | 12.2.1 | Display of adverse events | 47 |
| 1. | 2.3 | Serious Adverse Events and deaths. | 49 |
| | 12.3.1 | Serious Adverse Events | 49 |
| | 12.3.2 | Deaths | 50 |
| 1. | 2.4 | Clinical laboratory evaluation | 50 |
| | 12.4.1 | Hematological abnormalities | 50 |
| | 12.4.2 | Biochemical abnormalities | 52 |
| | 12.4.3 | Other metabolic parameters | 53 |
| | 12.4.4 | Laboratory values over time | 54 |
| 1. | 2.5 | Vital signs, physical findings, LVEF, ECG and other tests related to safety | 55 |
| | 12.5.1 | Vital signs and physical findings | 55 |
| | 12.5.2 | LVEF, ECG and other related tests | 55 |
| 1. | 2.6 | Concomitant therapy / procedures according to the ATC classification. | 56 |
| 1. | 2.7 | Safety analysis in special subgroups. | 57 |
| 13 | DB List | ings | 59 |
| 14 | Section | 16.2 ICH Listings | 60 |
| 15 | Referen | ces | 61 |

# ABBREVIATIONS AND GLOSSARY

| | Advance Front(c) |
|---|---|
| AE(s) | Adverse Event(s) |
| ALT | Angioimmunoblastic T-cell Lymphoma |
| ALT | All aline Aminotransferase |
| ALP | Alkaline Phosphatase |
| ASCT | Autologous Stem Cell Transplantation |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BL | Baseline |
| BMI | Body Mass Index |
| BSA | Body Surface Area |
| CI | Confidence Interval |
| CPK | Creatine Phosphokinase |
| CPK-MB | Serum CPK Isoenzymes (Found In Cardiac Muscle) |
| CR | Complete Remission |
| CRF | Case Report Form |
| CTCAE | National Cancer Institute Common Terminology Criteria for Adverse Events |
| DB | Data Base |
| DF | Degrees of Freedom |
| DoR | Duration of Response |
| ECG | Electrocardiogram |
| ЕСНО | Echocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| EOT | End of Treatment |
| EPO | Erythropoietin |
| FDA | Food and Drug Administration |
| FU | Follow-up |
| G-CSF | Granulocyte Colony Stimulating Factor |
| IA | Investigator Assessment |
| IDMC | Independent Data Monitorin Committe |
| Ig | Immunoglobulin |
| IPI | International Prognostic Index |
| IR | Independent Review |
| IRC | Independent Review Committee |
| LDH | Lactate Dehydrogenase |
| LVEF | Left Ventricular Ejection Fraction |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MUGA | Multiple-gated Acquisition Scan |
| NA | Not Applicable |
| | <u> </u> |
| NCI-CTCAE<br>NE | National Cancer Institute Common Terminology Criteria for Adverse Events Not Evaluable |
| | <u> </u> |
| NHL<br>NOS | Non-Hodgkin Lymphoma |
| | Not Otherwise Specified |
| ORR | Overall Response Rate |
| OS | Overall Survival |
| OS6 | Overall Survival at 6 months |
| OS12 | Overall Survival at 12 months |
| PCTL | Peripheral T-cell Lymphoma |
| PD | Progressive Disease |
| PFS | Progression-free Survival |
| PFS6 | Progression-free Survival at 6 months |
| PFS12 | Progression-free Survival at 12 months |
| PIAI | Prognostic Index for AITL |
| PIT | Prognostic Index for Peripheral T-cell lymphoma |

| PK | Pharmacokinetics |
|--------|-------------------------------------|
| PR | Partial Remission |
| PS | Performance Status |
| RBC | Red Blood Cell |
| R/R | Relapsed/Refractory |
| SAE(s) | Serious Adverse Event(s) |
| SD | Stable Disease |
| SOC | System Organ Class |
| SPD | Sum of the Product of the Diameters |
| StD | Standard Deviation |
| TTP | Time to Tumor Progression |
| ULN | Upper Limit of Normal |
| V | Version |
| WBC | White Blood Cells |
| WHO | World Health Organization |
| wk | Week |

#### 1 STUDY RATIONALE

Angioimmunoblastic T-cell lymphoma (AITL) is the second most common form of peripheral T-cell lymphoma (PTCL), accounting for approximately 20% of PTCLs and 2% of non-Hodgkin lymphomas (NHL). In the United States, the incidence is approximately 0.05 cases per 100,000 person years. The disease is more common in Europe (29% of PTCL cases) than in the United States or Asia.

The clinical course of AITL varies, with occasional spontaneous remissions. Nevertheless, the prognosis of the disease is dismal, with median survival < 3 years, and with 20–30% of long-term survivors. Different clinical risk factors as well as biological parameters have been described as prognostic factors. In a retrospective study of 157 cases of AITL, a multivariate analysis showed the following covariates as adversely associated with prognosis: male gender, anemia and the presence of mediastinal lymphadenopathy.

Other systems such as the International Prognostic Index (IPI) or the prognostic index for peripheral T-cell lymphoma (PIT) were of limited value in this disease. Recently, a risk model for AITL (prognostic index for AITL, PIAI) was designed based on the following adverse covariates: age > 60 years, performance status  $\ge 2$ , extranodal sites > 1, B-symptoms, and platelet count < 150,000/mL. The simplified PIAI had a low-risk group (zero to one factors) with a 5-year survival of 44%, and a high-risk group (two to five factors) with a 5-year survival of 24%.

In phase I studies conducted with plitidepsin, the schedule consisting of 1-hour i.v. infusion given weekly on D1, 8 and 15 q4wk was found to be the most convenient for patients with NHL. An exploratory phase II clinical trial (APL-B-013-02) was conducted to evaluate the efficacy, tolerability and pharmacokinetics of this weekly plitidepsin schedule at a starting dose of 3.2 mg/m² in patients with relapsed/refractory (R/R) aggressive NHL. This phase II trial included two cohorts: patients with non-cutaneous PTCL and patients with other aggressive lymphomas. No remissions were found in the cohort of 33 patients with other aggressive lymphomas. However, interesting antitumor activity was observed in 29 evaluable patients from the non-cutaneous PTCL cohort: ORR was 20.7% (95% CI, 8.0–39.7%) and SD rate was 20.7%.

Plitidepsin was well tolerated in this trial. The most common adverse events (AEs) in the non-cutaneous PTCL cohort were nausea, fatigue, vomiting, myalgia, muscle weakness and pyrexia. The most common grade 3/4 hematological abnormalities were lymphopenia, neutropenia, anemia and thrombocytopenia found in 28%, 12%, 10% and 10% of the cases, respectively.

Nine patients with AITL were included in the cohort of 34 non-cutaneous PTCL patients. Of note, ORR in these nine patients was 33.3%, with CR in two patients (22.2%) and PR in one patient (11.1%). Furthermore, SD was reported in other two patients. The median number of previous lines was 2 and the DoR of the three responders was 121, 12 and 4 weeks, respectively. It should be highlighted that the two patients with CR had bone marrow involvement at diagnosis and had previously failed high dose chemotherapy with stem cell transplantation (SCT) support.

In summary, the interesting antitumor activity observed with plitidepsin in non-cutaneous PTCL was mainly found in patients with AITL. Bearing in mind the small number of

agents with meaningful activity in non-cutaneous PTCL and, in particular, the lack of specific agents with reliable and specific activity in AITL, and considering the important signs of activity of plitidepsin in this disease, this phase II clinical trial was designed to evaluate plitidepsin as single-agent treatment for patients with R/R AITL.

The rationale of the exploratory biomarker objectives is related to recent studies exploring the genetic basis of the disease: a study by Odejide and colleagues showed high incidences of gene mutations of TET2, for example, in 85 AITL tissue samples, as well as in DNMT3A, and IDH2: common and frequent mutations that make AITL more comparable to myeloid disorders than other PTCLs and suggest the need to re-evaluate therapeutic strategies.

Several studies have shown that plitidepsin induces apoptosis in a cell type- and dose-dependent manner, and these effects are related to the induction of early oxidative stress, the activation of Rac1 GTPase and the inhibition of protein phosphatases, which in conjunction cause the sustained activation of JNK and p38 MAPK. The final consequence is the triggering of the mitochondrial apoptotic pathway with caspase 9 and caspase 3 activation. Additional effects may be mediated by indirect effects on the cell microenvironment, mainly mediated by antiangiogenic properties and indirect effects on monocyte-derived cells, including follicular dendritic cells.

## 2 STUDY DESIGN

Prospective, multicenter, phase II clinical trial.

The aim of this clinical trial is to determine the efficacy of plitidepsin in patients with relapsed/refractory AITL. A total of 60 patients will receive plitidepsin. The primary endpoint will be the ORR according to the Lugano classification response criteria per independent central review.

An Independent Review Committee (IRC) consisting of medical specialists (radiologists and hematologists) who are directly involved in the care of patients with AITL but do not take part in this trial as investigators or sub-investigators, will review all efficacy data and will assign the date of objective response or progression/censoring according to their independent evaluation.

Two futility analyses of the primary endpoint (ORR according to Lugano classification response criteria and per IRC) are planned around six months after approximately 25% and 50% of eligible patients (i.e., 15 and 30 patients respectively with AITL confirmed by central pathological review) have been treated. Two or less responders out of 15 patients or seven or less responders out of 30 patients, according to boundaries and sample size assumptions, will mean that the alternative hypothesis could be rejected, and thus recruitment might be stopped at the time of the first or second futility analysis, respectively. Otherwise, accrual will continue to a total of 60 patients with AITL confirmed by central pathological review. This decision will be taken at the time by an Independent Data Monitoring Committee (IDMC). The IDMC, which will include specialists in PTCL supported by a medical statistician, will review data provided by the Investigators, the IRC efficacy assessments and safety information and will advise whether the study should continue. Recruitment can continue during the review period.

If there are 19 or more responders over the total of 60 patients, the efficacy of plitidepsin will be considered as clinically relevant in AITL patients.

Operational details for the IRC and IDMC will be detailed in the corresponding charters.

## 3 OBJECTIVES AND ENDPOINTS

## 3.1 Primary objective

• To evaluate the efficacy of plitidepsin on the basis of overall response rate (ORR) in patients with relapsing/refractory angioimmunoblastic T-cell lymphoma (AITL).

## 3.2 Secondary objectives

- To evaluate other efficacy endpoints (time-to-event parameters: duration of response [DoR], progression-free survival [PFS], PFS at 6/12 months [PFS6/PFS12], intrapatient PFS/TTP, overall survival [OS] and OS at 6/12 months [OS6/OS12]).
- To evaluate the safety profile of plitidepsin in this patient population.
- To characterize the pharmacokinetics (PK) of plitidepsin.
- To identify biomarkers that may be predictive of plitidepsin activity.

## 3.3 Endpoints

# Primary endpoint:

• Overall response rate (ORR), defined as the percentage of patients with remission, either complete (CR) or partial remission (PR), according to the Lugano classification response criteria per independent central review. An external IRC will assign the objective response and a progression or censoring date for each patient.

### Secondary endpoints:

- ORR per investigator.
- CR rate, defined as the percentage of patients with complete remission according to the Lugano classification response criteria per independent central review and investigator assessment.
- Duration of response (DoR), defined as the time from the date when the remission criteria (PR or CR, whichever is first achieved) are fulfilled to the first date when PD, recurrence or death (due to any cause) is documented. Response will be assessed according to the Lugano classification response criteria per independent central review and investigator assessment.
- Progression-free survival (PFS), defined as the time from the date of first drug administration to the date of PD, death (of any cause), or last tumor evaluation; both independent central review and investigator assessment will be used for the determination of PFS.

- Progression-free survival at 6/12 months (PFS6/PFS12), defined as the Kaplan-Meier estimate of the percentage of patients who are progression-free at six/twelve months after first drug administration; both independent central review and investigator assessment will be used for the determination of PFS.
- Intrapatient PFS/TTP, defined as the ratio of PFS achieved with the experimental treatment *versus* the prior last TTP in the R/R setting.
- Overall survival (OS), defined as the time from the date of first dose to the date of death (of any cause) or last patient contact.
- Overall survival at 6/12 months (OS6/OS12), defined as the Kaplan-Meier estimate of the percentage of patients who are live at six/twelve months after first drug administration.
- Treatment safety [AEs, serious adverse events (SAEs) and laboratory abnormalities] graded according to the NCI-CTCAE, v. 4. Dose reductions, skipped doses or dose delays required due to treatment-related AEs, and reasons for treatment discontinuations will be analyzed.
- <u>Pharmacokinetics (PK)</u>, samples for PK analysis will be obtained during Cycle 1 exclusively.
- Exploratory biomarker analysis, correlation of efficacy with molecular markers (targets/pathways) related to the mechanism of action of plitidepsin or to the disease.

## 4 PATIENTS EVALUABILITY CRITERIA

The study population will include patients who have relapsed or refractory AITL confirmed by local pathological assessment. To be included in this study, the patients must meet all inclusion criteria and no exclusion criteria.

## 4.1 Analysis sets definitions

"All Included Patients" analysis set is defined as all patients who are included in the study (excluding patients who signed informed consent but are classified as screening failures), independent of whether they received the study drug.

"All Treated Patients" analysis set is defined as all included patients who receive at least part of one dose or infusion of plitidepsin.

"Per Protocol Patients" analysis set is defined as all eligible and treated patients with AITL diagnosis confirmed after central pathological review.

"All Evaluable Patients" analysis set is define as all eligible patients with AITL diagnosis confirmed after central pathological review who receive at least two plitidepsin cycles in which at least two complete infusions have been administered and had at least one disease assessment as well as in patients who discontinue treatment without Cycle 3 tumor assessment after at least two plitidepsin infusions due to disease progression (PD) (or death due to PD) or toxicity (or death due to toxicity), defined as "early PD" and "treatment failures" respectively.

"All Responder Patients" analysis set is defined as all patients with CR or PR as overall best response.

# 4.2 Efficacy populations

The "All Included Patients" analysis set will be used to show demographic and other baseline characteristics.

The "Per Protocol Patients" analysis set will be used for the primary endpoint analysis of ORR by IRC and for the secondary analyses of ORR by investigator assessment, CR rate and PFS analyses, as well as for OS analyses.

The "All Evaluable Patients" and "All Treated Patients" analysis sets will be used for the secondary endpoint analyses of ORR by IRC, ORR by investigator assessment, CR rate and PFS analyses, as well as for OS analyses.

The "All Responder Patients" dataset will be used for the duration of response (DoR) calculation

# 4.3 Safety population

The safety analysis is based on the "All Treated Patients" analysis set.

#### 5 SAMPLE CONSIDERATIONS

The primary endpoint for this study is ORR according to the Lugano classification response criteria per independent review in "Per Protocol Patients" population.

A total of 60 patients with AITL confirmed by central pathological review will be treated, 19 or more responders will be needed to get an overall estimate for response rate higher than 30% and its lower limit for the 95% confidence interval greater than 20% (31.7% CI95% 20.3%–45.0% following the binomial distribution).

The type I error (alpha) associated with this one-sided test is 0.025 and the type II error (beta) is 0.1; hence, statistical power is 90%. The null hypothesis (H0) is set at  $ORR \le 20\%$  (P0=0.208) versus the alternative hypothesis (H1) at  $\ge 40\%$  patients (Pa=0.41) having an objective response, the variance of the standardized test is under the null hypothesis.

Two futility analyses of the primary endpoint (ORR according to Lugano classification and per IRC) are planned to reject the alternative hypothesis six months after 25% and 50% of eligible patients have been treated (15 and 30 patients, respectively). Pocock boundary and the actual number of patients confirmed by central pathological review will be used to control type II error for both analyses. For example, if there are two or less responders out of 15 patients or seven or less responders out of 30 patients, according to boundaries and sample size assumptions, the alternative hypothesis could be rejected, and thus recruitment might be stopped at the time of the first or second futility analysis, respectively. Otherwise,

accrual will continue to a total of 60 patients AITL confirmed by central pathological review. Active recruitment will not be halted while the analysis is being carried out.

Therefore, if there are 19 or more responders of 60 patients, the null hypothesis can be rejected, allowing consideration of the observed activity plitidepsin as clinically relevant in the setting of patients with AITL.

## 6 STATISTICAL METHODOLOGY FOR EFFICACY

# 6.1 Planned analyses and definitions

## 6.1.1 Primary endpoint analysis

**Objective response** is defined as having partial remission (PR) or better as best overall response based on the Lugano classification response criteria per independent review. The **objective response rate (ORR)** is calculated as the number of objective responders divided by the number of patients in the "Per Protocol Patients" analysis set.

## 6.1.2 Secondary endpoints analyses

The *overall response rate (ORR)* is calculated as the number of objective responders based on the Lugano classification response criteria per independent review divided by the number of patients in the "All Evaluable Patients" and "All Treated Patients" analysis sets.

The *overall response rate (ORR)* is calculated as the number of objective responders based on the investigator criteria divided by the number of patients in the "Per Protocol Patients", "All Evaluable Patients" and "All Treated Patients" analysis sets.

The *complete remission rate* is calculated as the number of patients with complete remission based on the Lugano classification response criteria per independent review or per investigator assessment divided by the number of patients in the "Per Protocol Patients", "All Evaluable Patients" and "All Treated Patients" analysis sets.

The *duration of response (DoR)* will be analyzed in the "All Responder Patient". Duration of response will be calculated from the date of first documentation of response to the date of disease progression, recurrence or death with the same censoring rules as PFS. Response will be assessed according to the Lugano classification response criteria per independent central review and investigator assessment.

**Progression-free survival (PFS)** is defined as the time from the date of first administration to the date of documented progressive disease (PD) or death (regardless of the cause of death). If the patient receives further antitumor therapy (including stem cell transplant) before, PFS will be censored on the date of the last disease assessment prior to the administration of this antitumor therapy. If the patient is lost to follow-up for the assessment of progression the PFS will be censored at the date of last valid tumor assessment. If the patient does not received any drug infusion, he/she will be censored at time zero. Both, independent central review and investigator assessments, will be used for the determination of PFS.

**Progression-free survival at 6/12 months (PFS6/PFS12)**, defined as the Kaplan-Meier estimate of the percentage of patients who are progression-free at six/twelve months after first administration; both independent central review and investigator assessment will be used for the determination of PFS.

Within-patient PFS/TTP, defined as the ratio of the PFS achieved with the experimental treatment versus prior last TTP. Intra-patient PFS/TTP ratio will be categorized and analyzed as a dichotomous variable. Clinical benefit will be defined if a >33% longer PFS/TTP with the experimental treatment vs. the TTP with the immediate prior chemotherapy (ratio >1.33) is achieved.

Overall survival (OS), defined as the time from the date of first administration to the date of death (of any cause) or last patient contact.

*Overall survival at 6/12 months (OS6/OS12)*, defined as the Kaplan-Meier estimate of the percentage of patients who are alive at six/twelve months after first administration.

**Treatment safety** [AEs, serious adverse events (SAEs) and laboratory abnormalities] graded according to the NCI-CTCAE, v. 4. Dose reductions, skipped doses or dose delays required due to treatment-related AEs, and reasons for treatment discontinuations will be analyzed.

### 6.2 Efficacy analysis methods

# 6.2.1 Primary endpoint

For the evaluation of the main primary endpoint, *ORR*, the "Per Protocol Patients" population, the data from the Independent Review will be used. Binomial estimates with exact 95% CIs will be calculated for the analysis of response rate. A supportive analysis will be also done in the "All Evaluable Patients" and "All Treated Patients" populations and by investigator assessment as a secondary analysis.

#### 6.2.2 Secondary analyses

Time to event endpoints will be used in an exploratory way.

Binomial estimates with exact 95% CIs will be calculated for the analysis of *complete remission rate* in the "Per Protocol Patients", "All Evaluable Patients" and "All Treated Patients" analysis sets by independent review and investigator assessment.

**Duration of response** will be analyzed according to the Kaplan-Meier method in "All Responder Patients" analysis set by independent review and investigator assessment.

*Time to response* id defined as the time, in months, from the date of first drug administration to the first documentation of response method in "All Responder Patients" analysis set by independent review and investigator assessment.

**PFS** analysis will be performed in "Per Protocol Patients", "All Evaluable Patients" and "All Treated Patients" analysis sets according to the Kaplan-Meier method by independent review and investigator assessment. The concordance between the IRC and investigator evaluation of response and PFS will be shown using counts and percentages.

**OS** analysis will be performed in "Per Protocol Patients", "All Evaluable Patients" and "All Treated Patients" analysis sets according to the Kaplan-Meier.

Univariate evaluation of the influence of different prognostic factors on the main efficacy endpoints will be performed. If appropriate, univariate analyses will include prognostic factors/covariates widely reported and recognized by hematologist such as: sex, age at diagnosis, baseline ECOG, Body Surface Area, Ann arbor, extranodal disease, bone marrow involvement, B symptoms, baseline LDH xULN, bulky lesion, IPI, PIT, PIAI, Relapse or refractory, number of prior lines of treatment, previous SCT or time from last PD before inclusion. Further covariates could be included upon hematologist criteria. . . . . .

Cox proportional hazard models for PFS and OS, and logistic regression models for ORR will include the prognostic factors specified for the univariate analysis. More relevant and explanatory covariates from the univariate analysis will be included in the multivariate analyses (p-value < 0.10). Prognostic factors with more than 10% missing values will be excluded in the multivariate analyses.

### 7 STATISTICAL METHODOLOGY FOR SAFETY

Patients are evaluable for general safety if they received any study treatment.

### 7.1 Toxicity and adverse events

All the adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

The toxicity evaluation will be coded with the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.

As far as all the toxicities are concerned, the NCI-CTCAE grade will be used wherever an NCI-CTCAE grading exists. Otherwise, the severity will be noted. As a convention, the term «Grade» will always be used. Toxicities will be described according to the worst NCI-CTCAE grade or, for toxicities which do not form the subject of NCI-CTCAE classification, according to the worst severity. For "Worst per cycle" calculation purpose, onset and end cycle of each event will be derived.

Summary of overall adverse events will be done by body system and preferred term, by severity (worst toxicity grade) and by relationship to the study drug. Events with unknown relationship will be considered as related events for reporting purposes.

A frequency table will be made for the AEs leading to cycle delay, dose reduction, skipped dose, or withdrawal of study medication. Adverse events with outcome of death will also be presented by relationship to the study drug.

All events entered in Adverse Event form with the onset date before the first drug administration, will be reported as Signs and symptoms. Only those events with start date after/equal the first infusion date will be included in AE tables in Safety section (except those including evolution from baseline).

# 7.2 Clinical laboratory evaluation

Laboratory results will be classified according to the NCI-CTCAE version 4. All laboratory visits reported as "End of treatment" visit will be mapped to the last cycle visit.

For hematology values: absolute neutrophil count, lymphocyte count, WBC count, platelet count and hemoglobin worst grade per patient and per cycle will be displayed.

Time and duration of anemia, neutropenia and thrombocytopenia in cycles with grade 3-4 abnormality will be tabulated.

Overall cross tabulation will be presented for the worst grade during treatment versus the baseline toxicity grading of anemia, lymphopenia, leukopenia, neutropenia and thrombocytopenia.

The worst grade per patient during treatment and per cycle will be also calculated for the biochemical tests: ALT, AST, Total bilirubin, AP, CPK, creatinine, calcium, potassium, sodium, glucose and albumin.

Time and duration of AST, ALT and CPK increases in cycles with grade 3-4 abnormality will be tabulated.

Overall cross tabulation will be presented for the worst grade during treatment versus the baseline toxicity grading of AST, ALT and CPK increase.

# 7.3 Vital signs, physical examination, left ventricular ejection fraction (LVEF) and electrocardiogram findings

Tabulation will be made summarizing the performance status, body weight, LVEF and electrocardiogram abnormalities at baseline and during the treatment for each patient.

#### 7.4 Deaths and other Serious Adverse Events

Deaths and other Serious Adverse Events will be tabulated.

## 8 OTHER ANALYSES

Non-continuous variables will be described in frequency tables using counts and percentages. Continuous variables will be described by median, mean, standard deviation, minimum and maximum.

## 8.1 Baseline and demographic data

Baseline data such as demographics, disease history, prior therapy, prior relevant history, signs and symptoms, electrocardiogram, LVEF, protein measurements, laboratory values and concomitant medication (ATC-WHO coded) will be described following standard tables detailed in Appendix I. When two or more assessments have been done for the same parameter, the last assessment before or on the first drug administration will be taken into account for the analysis.

#### 8.2 Treatment administration

CRF cycles with a theoretical duration of 4 weeks will be used for this analysis.

Total cumulative dose, time on treatment, dose intensity and relative dose intensity, cycle delay, dose omissions, and dose reductions will be described following standard tables detailed in Appendix I.

Total cumulative dose, expressed in mg/m<sup>2</sup> is the sum of all the plitidepsin doses from the first cycle until last cycle including the dose received in last cycle.

Patients will be considered to be on-treatment for the duration of their treatment and 30 days following the last treatment dose. If the patient starts any new antitumor therapy outside this clinical trial or dies within 30 days of last treatment dose, the date of administration of this new therapy or the date of death will be considered the date of treatment discontinuation.

However, as a convention, for dose intensity calculation purposes, the duration of the last cycle is considered to be 28 days.

Intended dose intensity is the planned dose per cycle divided by the planned number of weeks by cycle (2.4mg/m²/wk for plitidepsin).

Absolute dose intensity is the actual cumulative dose divided by the number of weeks of treatment. Relative dose intensity (%) is the ratio of absolute dose intensity divided by the intended dose intensity.

The item «Infusion delayed: yes/no» in the case report form (CRF) will be used to calculate the delay (on day 1 infusion). For cycles considered as delayed by the investigator, the delay will be calculated as:

Delay: Date of current drug administration – Date of previous drug administration – 28.

The first infusion of the first cycle will be excluded from all cycle delay and cycle modification calculations.

#### 8.3 Subsequent therapy

A table summarizing the subsequent therapies received after treatment discontinuation will be shown

Time to first subsequent therapy or death will be analyzed as a measure of the time from first drug administration to treatment failure that leads to the need of a further treatment regimen.

#### 8.4 Protocol deviations

Analysis of inclusion/exclusion criteria deviations, retreatment restrictions, used concomitant medication and clinically relevant discontinuations will be done as described in Appendix I.

#### 8.5 Pharmacokinetic and biomarkers analyses

These analyses will be detailed in separate documents.

# 8.6 Imputation of incomplete dates

The dates of certain historical or current clinical activities are key component for statistical analysis. Incomplete date appears when day, month or year is/are missing, and it could be imputed so that variables like time to and duration of certain event can be calculated. If none of day, month and year is available, then the date is missing, no imputation will be done.

## Before treatment start date

If day of a date is unknown then the imputed day will be 15, if the month is also unknown then the imputed date will be July 1st. This assumption will be valid if the imputed date is earlier than the treatment start date; otherwise the imputed date will be the first day of the treatment start month.

# Between treatment start and end of treatment

All date variables during treatment where information is needed and is not fully available, for example adverse events or concomitant medications, will be subject of imputation by means of SAS programming. If the day of a date is unknown then the imputed day will be 1, if the month and/or year is also unknown then the imputed date will 1/January. This assumption will be valid if the imputed date is earlier than the treatment start date; otherwise, the imputed date will be the treatment start date.

### After end of treatment

To ensure the most conservative approach for the main time-to-event variables (i.e. PFS and OS) that can be affected by missing values the following rules will be implemented by means of SAS programming: if the day of a date is unknown then the imputed day will be 1; if the month is also unknown, then the imputed date will be 1/July. This assumption will be valid if the imputed date occurs later than the last drug administration date; otherwise, the imputed date will be the last drug administration date plus 1 day.

#### 8.7 Subgroup analyses

No specific subgroup analysis is planned for efficacy. However, the influence of prognostic factors on the efficacy endpoints will be studied in the multivariate analysis.

No formal statistical allowance will be made for multiple subgroup investigations, but any apparent subgroup interactions will be interpreted appropriately in a cautious way.

Analysis of safety profile by age, gender, race and body mass index (BMI) will be provided as specified in section 12.7.

## Handling of multicenter data

Not applicable.

## Handling of multiple comparisons

No formal statistical allowance will be made for multiple comparisons, therefore any apparent subgroup analysis will be interpreted appropriately in a cautious way.

## 8.8 Decimal places and methods for handling missing data

By default, all results will be rounded to one decimal, except in the case where variables are integer; in that case, they will be reported without decimals, for example, age in years, number of sites. For representing p-values four decimals will be selected as default but they could be rounded to fewer decimals if necessary. Missing values will not be included in the calculation of outputs.

### 8.9 Interim and group sequential analyses

Two futility analyses of the primary endpoint (ORR according to the Lugano classification response criteria per independent review) are planned to reject the alternative hypothesis when  $\sim\!25\%$  and  $\sim\!50\%$  of the patients have been recruited (first 15 and 30 patients, respectively). Pocock boundary and the actual number of patients confirmed by central pathological review will be used to control type II error for both analyses. For example, if there are two or less responders out of 15 patients or seven or less responders out of 30 patients, according to boundaries and sample size assumptions, the alternative hypothesis could be rejected, and thus recruitment might be stopped at the time of the first or second futility analysis, respectively.

## 8.10 Identification of fixed or random effects models

Not applicable

#### 9 STATISTICAL SOFTWARE

Medidata Rave® EDC will be used for data entry and clinical data management. EAST v5.2 has been used to calculate sample size. SAS v9 (1) or superior will be used for all statistical analysis outputs.

#### APPENDIX I

All tables will be created at the time of each analysis planned in the protocol if applicable, and at study end.

# 10 Study Patients

These analyses will be performed in "All Included patients" analysis set.

# 10.1 Patient disposition

Main characteristics concerning inclusion in the study, withdrawal from the study and protocol deviations will be displayed in this section.

Table 10.1.1 Number of patients per population

| | N | % |
|------------------------|---|-----|
| All Included Patients | X | X.X |
| All Evaluable Patients | | |
| All Treated Patients | | |
| Per Protocol Patients | | |

Listing 10.1.2 Patients excluded from analysis populations

| Patient id. | Population | Exclusion reason |
|-------------|------------|------------------|

Table 10.1.3 Patients accrual by institution

| | Country | Institution | N | % |
|--------------|-----------|---------------|---|-----|
| | | Institution 1 | X | X.X |
| | Country 1 | | | |
| | | Total | | |
| | | Institution 1 | | |
| No. included | | | | |
| | | Total | | |
| | | Institution 1 | | |
| | Total | | | |
| | | Total | | |
| | | Institution 1 | | |
| | Country 1 | | | |
| | | Total | | |
| | | Institution 1 | | |
| No. treated | | | | |
| | | Total | | |
| | | Institution 1 | | |
| | Total | | | |
| | | Total | | |

# Table 10.1.4 Study dates

| racio rolli stady dates |
|-----------------------------------------|
| Date of first registration |
| Date of first dose of the first patient |
| Date of last registration |
| Date of first dose of the last patient |
| Date of last dose |
| Date of last follow-up* |

<sup>(\*)</sup> Last follow-up or exam or procedure before clinical cut-off or study closure

# 10.2 Reasons for treatment discontinuation

## Table 10.2.1 Treatment discontinuation

| | N | % |
|---|---|---|
| Progressive disease | X | X.X |
| Treatment related adverse event | | |
| Non treatment related adverse event | | |
| Patient refusal to treatment | | |
| Investigator decision | | |
| Death (due to toxicity)* | | |
| Death (non-treatment-related)** | | |
| Complete response | | |
| PR or CR and eligible for consolidation with autologous or allogeneic SCT | | |
| Other *** | | |
| Total | | |

<sup>(\*)</sup> Cause of death = study drug related (\*\*) Cause of death = Malignant disease / non study drug related / Other (\*\*\*) Specify (see listing 10.2.2). Patients included but not treated will not be shown in this table.

When reason for discontinuation is toxicity or study treatment-related death, identify patients and describe them in depth here.

Listing 10.2.2 Reasons for treatment discontinuation other than progressive disease.

| Patient id. | Reason | Last cycle | Comments |
|-------------|--------|------------|----------|

## Listing 10.2.3 Treatment discontinuation due to AEs

| Patient id. | Cycle | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset<br>date | Resolved date | Significant consequences |
|---|---|---|---|---|---|---|---|---|

# Table 10.2.4 Study discontinuation

| | | N | % |
|---|---|---|---|
| Study termination (clinical cut-off) | | X | X.X |
| Patient's refusal | | | |
| Never treated* | | | |
| Death (due to toxicity)** | | | |
| Death (non-treatment-related)*** | | | |
| Investigator decision | | | |
| Patient's follow-up completed | | | |
| Lost to follow-up | | | |
| Other **** | | | |
| Total | • | | |
| (d) G T' : 10 0 C (d) G C 1 1 . 1 1 1 . 1 (d) d) d) | G C1 1 | 3.6.12 | / . 1 1 |

<sup>(\*)</sup> See Listing 10.2.6 (\*\*) Cause of death = study drug related (\*\*\*) Cause of death = Malignant disease / non study drug related / Other (\*\*\*\*)See Listing 10.2.5

# Listing 10.2.5 Study discontinuation due to other reason

| Patient id. | Specify |
|-------------|---------|

### Listing 10.2.6 Patients included but not treated

| Patient id. | Off-study reason |
|-------------|------------------|

Listing 10.2.7 Patients included without AITL diagnosis confirmed after central pathological review

| p will be grown to vie vi | |
|---------------------------|---------------|
| Patient id. | Treated (Y/N) |

# 10.3 Protocol deviations

Listing 10.3.1 Protocol deviations

| Patient id. | Deviation type | Description |
|-------------|----------------|-------------|

# 11 Efficacy Evaluation

# 11.1 Demographic and other baseline characteristics

These analyses will be performed in "All Included patients" analysis set.

# 11.1.1 Patient characteristics at baseline

Table 11.1.1.1 Baseline characteristics: Gender

| | N | % |
|--------|---|-----|
| Male | X | X.X |
| Female | | |
| Total | | |

Table 11.1.1.2 Baseline characteristics: Age at treatment registration

| N | Median | Mean | StD | Min | Max |
|---|--------|------|-----|-----|-----|

Table 11.1.1.3 Baseline characteristics: Age grouped

| | N | % |
|-------|---|-----|
| 18-XX | X | X.X |
| XX-YY | | |
| ≥65 | | |
| Total | | |

# Table 11.1.1.4 Baseline characteristics: Race

| | N | % |
|-------|---|-----|
| White | X | X.X |
| Total | | |

# 11.1.2 Local histopathological diagnosis

# Table 11.1.2.1 Histopathological diagnosis: Clinical features

| Systemic clinical manifestations | N | % |
|-----------------------------------|---|-----|
| Generalized lymphadenopathy | X | X.X |
| Hepatosplenomegaly | | |
| Skin rash/pruritus | | |
| Polyclonal hypergammaglobulinemia | | |
| Others | | |

# Listing 11.1.2.2 Histopathological diagnosis: Clinical features, other clinical manifestations

| Patient id. | Other systemic clinical manifestations |
|-------------|----------------------------------------|

Table 11.1.2.3 Histopathological diagnosis: Pathologic and immunophenotypic features

| | <u> </u> | 1 71 |
|---|---|---|
| Common T-cell markers (Positive) | N | % |
| CD3 | X | X.X |
| CD4 | | |
| CD8 | | |
| Other markers | | |
| Expression of follicular TH (TFH) markers by the tumor cells | N | % |
| (Positive) | | |
| PD1 | X | X.X |
| BCL6 | | |
| CXCL13 | | |
| CD10 | | |
| ICOS | | |
| Hyperplasia of follicular dendritic cells (CD23+ and/or CD21+) | N | % |
| Hyperplasia of follicular dendritic cells (Present) | X | X.X |
| EBV in-situ hybridization (EBERs) (Positive) | | |
| Presence of CD30+ B-cell blast (Positive) | | |
| Other relevant features | | |

Listing 11.1.2.4 Histopathological diagnosis: Other common T-cell markers

| Patient id. | Other common T-cell markers |
|-------------|-----------------------------|

# Listing 11.1.2.5 Histopathological diagnosis: Other relevant hyperplasia of follicular dentritic cell features

| Patient id. | Other relevant features |
|-------------|-------------------------|

# Listing 11.1.2.6 Patients without AITL diagnosis confirmed by local histopathological report

| Patient id. | Reason |
|-------------|--------|

# 11.1.3 Disease at diagnosis, time from diagnosis and current disease

Table 11.1.3.1 Time from diagnosis to first infusion (months)

| N | Median | Mean | StD | Min | Max |
|---|--------|------|-----|-----|-----|
| X | X.X | X.X | X.X | X.X | X.X |

# Table 11.1.3.2 Time from last PD\* to first infusion (weeks)

| N | 1 | Median | Mean | StD | Min | Max |
|---|---|--------|------|-----|-----|-----|
| X | | X.X | X.X | X.X | X.X | X.X |

<sup>(\*)</sup>PD date will be taken from Lymphoma History form as date of relapsed or refractory disease. If the day or the month or the full date is missing, further information will be taken from Prior anticancer therapy form. After that, if the date is still incomplete, imputation rules described in section 8.6 will be used.

| Table 11.1.3.3 | A mm A mhan | I v maa mala a maa a | ata a a at | diamagia |
|----------------|-------------|----------------------|------------|----------|
| Table III 7 7 | AIIII-AIDOI | LAHIDHOHIA | STAGE AL | HAVIOSIS |

| | N | % |
|-------|---|-----|
| I-A | X | X.X |
| I-B | | |
| II-A | | |
| Total | | |

# Table 11.1.3.4 Ann-Arbor Lymphoma stage at diagnosis I/II vs III/IV.

| | N | % |
|--------|---|-----|
| I/II | X | X.X |
| III/IV | | |
| Total | | |

# Table 11.1.3.5 Extranodal disease at diagnosis.

| | N | % |
|-------|---|-----|
| Yes | X | X.X |
| No | | |
| Total | | |

# Listing 11.1.2.6 Extranodal sites at diagnosis.

| Patient id. | Extranodal sites |
|-------------|------------------|

# Table 11.1.3.6 Bulky lesion at diagnosis

| | N | 0% |
|-------|---|------|
| Yes | X | XX.X |
| No | | |
| Total | | |

# Table 11.1.3.7 International Prognostic Index at diagnosis

| | N | % |
|-----------------------------------------|---|-----|
| Low risk (0-1 risk factors) | X | X.X |
| Low-intermedite risk (2 risk factors) | | |
| High-intermediate risk (3 risk factors) | | |
| High risk (4-5 risk factors) | | |
| Not available | | |
| Total | | |

# Table 11.1.3.8 Prognostic Index for Peripheral T-Cell Lymphoma (PIT) at diagnosis

| | N | % |
|---------------|---|-----|
| Group 1 | X | X.X |
| Group 2 | | |
| Group 3 | | |
| Group 4 | | |
| Not available | | |
| Total | | |

# Table 11.1.3.9 Prognostic Index for Angioimmunoblastic T-Cell Lymphoma (PIAI) at diagnosis

| $\mathcal{E}$ | | |
|-----------------|---|-----|
| | N | % |
| Low risk group | X | X.X |
| High risk group | | |
| Not available | | |
| Total | | |

# Table 11.1.3.10 Relapsed / Refractory at current disease

| | N | % |
|------------|---|-----|
| Relapsed | X | X.X |
| Refractory | | |
| Total | | |

# Table 11.1.3.11 International Prognostic Index at current disease

| | N | % |
|-----------------------------------------|---|-----|
| Low risk (0-1 risk factors) | X | X.X |
| Low-intermedite risk (2 risk factors) | | |
| High-intermediate risk (3 risk factors) | | |
| High risk (4-5 risk factors) | | |
| Not available | | |
| Total | | |

# Table 11.1.3.12 Prognostic Index for Peripheral T-Cell Lymphoma (PIT) at current disease

| | N | % |
|---------------|---|-----|
| Group 1 | X | X.X |
| Group 2 | | |
| Group 3 | | |
| Group 4 | | |
| Not available | | |
| Total | | |

# Table 11.1.3.13 Prognostic Index for Angioimmunoblastic T-Cell Lymphoma (PIAI) at current disease

| | N | % |
|-----------------|---|-----|
| Low risk group | X | X.X |
| High risk group | | |
| Not available | | |
| Total | | |

# Table 11.1.3.14 Baseline characteristics: protein measurements

| | N | Median | Mean | StD | Min | Max |
|-------------|---|--------|------|-----|-----|-----|
| Ig G (g/dl) | X | X.X | X.X | X.X | X.X | X.X |
| Ig A (g/dl) | | | | | | |
| Ig M (g/dl) | | | | | | |

## Listing 11.1.3.15 Baseline characteristics: protein measurements

| Patient id. | Date | Ig G (g/dl) | Ig A (g/dl) | Ig M (g/dl) | Immunofixation serum |
|---|---|---|---|---|---|

# 11.1.4 Prior anticancer therapy

Listing 11.1.4.1 Patients with prior radiotherapy

| Patient id. | Intention | Site (Anatomic) | Total dose (Gy) | First dose | Last dose |
|---|---|---|---|---|---|

Listing 11.1.4.2 Patients with prior surgery

| Patient id. | Site and procedures | Date |
|-------------|---------------------|------|

Table 11.1.4.3 Number of lines of prior medical therapy

| | N | % |
|----------------|---|-----|
| 1 | X | X.X |
| 2 | | |
| Total | | |
| Median (Range) | | |

Table 11.1.4.4 Prior anticancer agents

| Antineoplastic and Immunomodulating agents (ATC-class.) | | |
|---------------------------------------------------------|---|-----|
| | N | % |
| Antineoplastic Agents (L01) | X | X.X |

Table 11.1.4.5 TTP to last prior anticancer therapy

| Time to progression. Last | N | Median | Mean | StD | Min | Max |
|-----------------------------|---|--------|------|-----|-----|-----|
| anticancer therapy (months) | | | | | | |
| Total | X | X.X | X.X | X.X | X.X | X.X |

Table 11.1.4.6 Response to last therapy

| | N | % |
|---------------|---|-----|
| CR | X | X.X |
| PR | | |
| SD | | |
| PD | | |
| NE / NA / UNK | | |

Table 11.1.4.7 Prior stem cell transplantation

| | N | % |
|------------|---|-----|
| 0 | X | X.X |
| 1 | | |
| ≥2 | | |
| Type | N | % |
| Autologous | X | X.X |
| Allogeneic | | |

# 11.1.5 Prior history

Listing 11.1.5.1 Prior history not resolved

| Patient id. | Description | Onset Date |
|-------------|-------------|------------|

# 11.1.6 Physical examination, vital signs, electrocardiogram and other tests

For the physical examination, vital signs, electrocardiogram and other tests, the last examination available before treatment will be described in the following tables.

Table 11.1.6.1 Baseline characteristics: Physical exam

| | N | % |
|-----------|---|-----|
| Normal | X | X.X |
| Abnormal* | | |
| Total | | |

(\*)See listing 11.1.6.2

# Listing 11.1.6.2 Physical examination abnormalities

| Patient id. | Body system examined | Onset Date |
|-------------|----------------------|------------|

## Table 11.1.6.3 Baseline characteristics: Physical exam and vital signs.

| Parameter | N | Median | Mean | StD | Min | Max |
|---------------------------------|---|--------|------|-----|-----|-----|
| Weight (kg.) | X | X.X | X.X | X.X | X.X | X.X |
| Height (cm.) | | | | | | |
| $BSA(m^2)$ | | | | | | |
| Heart rate (beats/min) | | | | | | |
| Systolic blood pressure (mmHg) | | | | | | |
| Diastolic blood pressure (mmHg) | | | | | | |
| Temperature (°C) | | | | | | |

# Table 11.1.6.4 Baseline characteristics: ECOG Performance Status

| | N | % |
|-------|---|-----|
| 0 | X | X.X |
| 1 | | |
| 2 | | |
| Total | | |

## Table 11.1.6.5 Baseline characteristics: Electrocardiogram

| | N | % |
|-------------------------------|---|-----|
| Normal | X | X.X |
| Significant abnormalities* | | |
| Non significant abnormalities | | |
| Total | | |

<sup>(\*)</sup>See tables of signs and symptoms or prior history for details and listing 11.1.6.6

# Listing 11.1.6.6 ECG abnormalities at baseline

| Patient id. | Result | Heart rate (bpm) | QT interval<br>(msec) | Fridericia<br>corrected QT<br>(msec) | Specify |
|---|---|---|---|---|---|

# Table 11.1.6.7 Baseline characteristics: LVEF

| | N | % |
|--------------------------------|---|-----|
| Normal | X | X.X |
| Significant abnormalities* | | |
| Non significant abnormalities* | | |
| Total | | |

<sup>(\*)</sup>See tables of signs and symptoms or prior history for details and listing 11.1.6.8

# Listing 11.1.6.8 Patients with Left Ventricular Ejection Fraction abnormalities at baseline

| | | | | , | |
|---|---|---|---|---|---|
| Patient id. | Date | Result | LVEF (%) | Institutional normal range (%) | Method |

# Table 11.1.6.9 Baseline characteristics Median and range of LVEF

| | N | Median | Mean | StD | Range |
|------|---|--------|------|-----|---------|
| MUGA | X | X.X | X.X | X.X | X.X-X.X |
| ЕСНО | | | | | |
| Both | | | | | |

Table 11.1.6.10 Baseline characteristics: Neurological examination

| | N | % |
|-----------|---|-----|
| Normal | X | X.X |
| Abnormal* | | |
| Total | | |

<sup>(\*)</sup>See tables of signs and symptoms or prior history for details and listing 11.1.6.11

Listing 11.1.6.11 Neurological examination abnormalities at baseline

| Patient id. | Result | Specify |
|-------------|--------|---------|

Table 11.1.6.12 Baseline characteristics: Urinary dipstick

| | N | % |
|-----------|---|-----|
| Normal | X | X.X |
| Abnormal* | | |
| Total | | |

<sup>(\*)</sup>See table 11.1.6.13 for further details

Listing 11.1.6.13 Patients with abnormal urinary dipstick at baseline

| Patient id. | Date | Result | Proteinuria | Leukocytes | Red Blood<br>Cells |
|-------------|------|--------|-------------|------------|--------------------|

## Table 11.1.6.14 Baseline characteristics: Coombs test result

| | N | % |
|----------|---|-----|
| Positive | X | X.X |
| Negative | | |
| Total | | |

Table 11.1.6.15 Baseline characteristics: Viral serology results

| | N | % |
|-----------------|---|-----|
| Hepatitis B | | |
| Positive | X | X.X |
| Negative | | |
| Not done | | |
| Total | | |
| Hepatitis C | | |
| Positive | X | X.X |
| Negative | | |
| Not done | | |
| Total | | |
| Cytomegalovirus | | |
| Positive | X | X.X |
| Negative | | |
| Not done | | |
| Total | | |

Listing 11.1.6.16 Patients with positive viral serology results at baseline

| Patient | | I | ) | Hepatitis C | Cyto | megalovirus | |
|---|---|---|---|---|---|---|---|
| | Date | Surface | Surface | Core antibody | HCV | CMV pp65 | Quantitative CMV |
| 1d. | | antigen | antibody | | | | DNA PCR |

Table 11.1.6.17 Baseline characteristics: Adequate contraception

| | N | % |
|-------|---|-----|
| Yes | X | X.X |
| No | | |
| NA* | | |
| Total | | |

<sup>(\*)</sup> Specify reasons

Table 11.1.6.18 Baseline characteristics: Pregnancy test

| | N | % |
|----------|---|-----|
| Yes | X | X.X |
| No | | |
| NA* | | |
| Not done | | |
| Total | | |

<sup>(\*)</sup> Specify reasons

# 11.1.7 Hematological values at baseline

Table 11.1.7.1 Hematological abnormalities at baseline

| | N | | ade<br>1 | <br>Gr | ade<br>4 | Al | 1* |
|------------------|---|---|----------|--------|----------|----|-----|
| | N | N | % | <br>N | % | N | % |
| Leukopenia | X | X | X.X | X | X.X | X | X.X |
| Anemia | | | | | | | |
| Thrombocytopenia | | | | | | | |
| Neutropenia | | | | | | | |
| Lymphopenia | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.7.2 Hematology values at baseline

| | N | Median | Mean | StD | Range |
|----------------------------------|---|--------|------|-----|---------|
| WBC $(10^9/L)$ | X | X.X | X.X | X.X | X.X-X.X |
| Hemoglobin (g/dL) | | | | | |
| Hematocrit (%) | | | | | |
| Platelets (10 <sup>9</sup> /L) | | | | | |
| Neutrophils (10 <sup>9</sup> /L) | | | | | |
| Lymphocytes (10 <sup>9</sup> /L) | | | | | |

Listing 11.1.7.3 Hematological tests not assessed at baseline

| Patient id. | Lab. test |
|-------------|-----------|

Listing 11.1.7.4 Hematological abnormalities at baseline. Grade > 2

| Patient id | Parameter | Value | Grade |
|------------|-----------|-------|-------|
| | | X X | |

# 11.1.8 Biochemical values at baseline

Table 11.1.8.1 Biochemical abnormalities at baseline

| | N | Grade<br>1 | | ••• | Grade<br>4 | | All* | |
|---|---|---|---|---|---|---|---|---|
| | N | N | % | | N | % | N | % |
| AST increase | X | X | X.X | | X | X.X | X | X.X |
| ALT increase | | | | | | | | |
| Total bilirubin increase | | | | | | | | |
| ALP increase | | | | | | | | |
| Creatinine increase | | | | | | | | |
| CPK increase | | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.8.2 Biochemical values at baseline

| | N | Median | Mean | StD | Range |
|-------------------------------|---|--------|------|-----|---------|
| AST (IU/L) | X | X.X | X.X | X.X | X.X-X.X |
| ALT (IU/L) | | | | | |
| Total bilirubin (mg/dL) | | | | | |
| Direct bilirubin (mg/dL) | | | | | |
| ALP (IU/L) | | | | | |
| Creatinine (mg/dL) | | | | | |
| Creatinine Clearance (ml/min) | | | | | |
| CPK (IU/L) | | | | | |
| CPK MB (IU/L) | | | | | |
| Total proteins (g/dL) | | | | | |
| Albumin (g/dL) | | | | | |
| Uric acid (mg/dL) | | | | | |
| LDH (IU/L) | | | | | |
| CRP (mg/dL) | | | | | |
| Beta-2-microglobulin (mg/L) | | | | | |

Listing 11.1.8.3 Biochemical tests not assessed at baseline

| Patient id. | | Lab. test |
|-------------|-----|-----------|
| | ••• | |

Listing 11.1.8.4 Biochemical abnormalities at baseline. Grade  $\geq 2$ 

| | | <del>_</del> | |
|------------|-----------|--------------|-------|
| Patient id | Parameter | Value | Grade |
| | | X.X | |

# 11.1.9 Other metabolic values at baseline

Table 11.1.9.1 Other metabolic abnormalities at baseline

| | N | Grade<br>1 | | <br>Grade<br>4 | | All* | |
|-----------------|---|------------|-----|----------------|-----|------|-----|
| | N | N | % | <br>N | % | N | % |
| Hyperglycemia | X | X | X.X | X | X.X | X | X.X |
| Hypoglycemia | | | | | | | |
| Hypoalbuminemia | | | | | | | |

<sup>(\*)</sup>Any grade

Table 11.1.9.2 Other metabolic values at baseline

| | N | Median | Mean | Std | Range |
|--------------------|---|--------|------|-----|---------|
| Sodium (mmol/L) | X | X.X | X.X | X.X | X.X-X.X |
| Potassium (mmol/L) | | | | | |
| Calcium (mmol/L) | | | | | |
| Magnesium (mmol/L) | | | | | |
| Glucose (mmol/L) | | | | | |

Listing 11.1.9.3 Metabolic tests not assessed at baseline

| Patient id. | Lab. test |
|-------------|-----------|

Listing 11.1.9.4 Metabolic abnormalities at baseline. Grade  $\geq 2$ 

| Patient id Parameter | Value | Grade |
|----------------------|-------|-------|
| | X,X | |

# 11.1.10 Signs and symptoms at baseline

Table 11.1.10.1 Patients with signs and symptoms at baseline

| <u> </u> | N | 0/2 |
|------------------------------------|-----------|-----|
| | 11 | /0 |
| No. signs and symptoms per patient | | |
| 0 | X | X.X |
| 1 | | |
| 2 | | |
| ≥ 3 | | |
| Median (Range) | X.X (X-X) | |

Table 11.1.10.2 Signs and symptoms at baseline

| | | N | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | N | % | <br>N | % | N | % |
| | | X | X | X.X | X | X.X | X | X.X |
| Gastrointestinal disorders | Diarrhea NOS | | | | | | | |
| General disorders and | Fatigue | | | | | | | |
| administration site conditions | | | | | | | | |

<sup>(\*)</sup>Any grade

Listing 11.1.10.3 Signs and Symptoms at baseline

| Patient id. | Sign/symptom | Grade | Onset date | Relationship | Treated |
|-------------|--------------|-------|------------|--------------|---------|

# 11.1.11 Concomitant therapy and procedures at baseline

Concomitant medication at baseline according to the ATC classification.

Table 11.1.11.1 Agents of concomitant therapy started at baseline

| Medication Term (ATC level 1) | Medication Term (ATC level 2) | Medication Term<br>(ATC level 4) | Preferred Name | N | % |
|---|---|---|---|---|---|
| | | | | X | X.X |

Listing 11.1.11.2 Concomitant therapy at baseline

| Patient id. | Туре | Drug name | ATC Code | Route | Total daily dose | Start date | Reason for use | Indication for therapeutic |
|---|---|---|---|---|---|---|---|---|
| 14. | | | | | 4050 | | | reason |

Listing 11.1.11.3 Concomitant procedures at baseline

| Patient id. | Procedure | Date | Indication | AE/MH/Other | Comments |
|-------------|-----------|------|------------|-------------|----------|

# 11.2 Measurements of treatment compliance

Not applicable.

# 11.3 Efficacy analysis

# 11.3.1 Primary analysis

Table 11.3.1.1 Response rate by the Lugano classification response criteria (Independent Review assessment and "Per Protocol Patients" population)

| Response | | |
|----------------|---|-----|
| | N | % |
| CR | X | X.X |
| PR | | |
| SD | | |
| CR PR SD PD NE | | |
| NE | | |

Table 11.3.1.2 Response rate estimates by the Lugano classification response criteria (Independent Review assessment and "Per Protocol Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------------|------------|-----------------|-----------------|
| Response rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.1.3 Response rate by the Lugano classification response criteria (Independent Review assessment and "Per Protocol Patients" population) in first futility analysis

| Response | N | % | Pocock |
|----------|---|-----|----------|
| | | | boundary |
| CR | X | X.X | |
| PR | | | |
| SD | | | |
| PD | | | |
| NE | | | |

Table 11.3.1.4 Response rate by the Lugano classification response criteria (Independent Review assessment and "Per Protocol Patients" population) in second futility analysis

| Response | N | % | Pocock |
|----------|---|-----|----------|
| | | | boundary |
| CR | X | X.X | |
| PR | | | |
| SD | | | |
| PD | | | |
| NE | | | |

# 11.3.2 Secondary analyses

Table 11.3.2.1 Response rate by the Lugano classification response criteria (Investigator assessment and "Per Protocol Patients" population)

| assessment and Territoteetri attents population) | | |
|--------------------------------------------------|---|-----|
| Response | | • |
| | N | % |
| CR | X | X.X |
| PR | | |
| SD | | |
| SD<br>PD<br>NE | | |
| NE | | |

Table 11.3.2.2 Response rate estimates by the Lugano classification response criteria (Investigator assessment and "Per Protocol Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------------|------------|-----------------|-----------------|
| Response rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.3 Response rate by the Lugano classification response criteria (Independent Review assessment and "All Evaluable Patients" population)

| Response | | |
|----------|---|-----|
| | N | % |
| CR | X | X.X |
| CR<br>PR | | |
| SD | | |
| PD<br>NE | | |
| NE | | |

Table 11.3.2.4 Response rate estimates by the Lugano classification response criteria (Independent Review assessment and "All Evaluable Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------------|------------|-----------------|-----------------|
| Response rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.5 Response rate by the Lugano classification response criteria (Investigator assessment and "All Evaluable Patients" population)

| assessment and 7 m Evaluable Lanents population) | | |
|--------------------------------------------------|---|-----|
| Response | | |
| | N | % |
| CR | X | X.X |
| PR | | |
| SD | | |
| PD | | |
| NE | | |

Table 11.3.2.6 Response rate estimates by the Lugano classification response criteria (Investigator assessment and "All Evaluable Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------------|------------|-----------------|-----------------|
| Response rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.7 Response rate by the Lugano classification response criteria (Independent Review assessment and "All Treated Patients" population)

| Response | | |
|----------------|---|-----|
| | N | % |
| CR | X | X.X |
| PR | | |
| SD | | |
| CR PR SD PD NE | | |
| NE | | |

Table 11.3.2.8 Response rate estimates by the Lugano classification response criteria (Independent Review assessment and "All Treated Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------------|------------|-----------------|-----------------|
| Response rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.9 Response rate by the Lugano classification response criteria (Investigator assessment and "All Treated Patients" population)

| Response | | |
|----------------------------|---|-----|
| | N | % |
| CR | X | X.X |
| PR | | |
| SD | | |
| CR<br>PR<br>SD<br>PD<br>NE | | |
| NE | | |

Table 11.3.2.10 Response rate estimates by the Lugano classification response criteria (Investigator assessment and "All Treated Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------------|------------|-----------------|-----------------|
| Response rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.11 ORR – Concordance between Independent Review assessment and Investigator assessment ("Per Protocol Patients" population)

| | | Response by Investigator assessment | | | |
|-----------------|----|-------------------------------------|----|----|----|
| Response by IRC | CR | PR | SD | PD | NE |
| CR | | | | | |
| PR | | | | | |
| SD | | | | | |
| PD | | | | | |
| NE | | | | | |

Table 11.3.2.12 CR rate estimates by the Lugano classification response criteria (Independent Review assessment and "Per Protocol Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------|------------|-----------------|-----------------|
| CR rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.13 CR rate estimates by the Lugano classification response criteria (Independent Review assessment and "All Evaluable Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------|------------|-----------------|-----------------|
| CR rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.14 CR rate estimates by the Lugano classification response criteria (Independent Review and "All Treated Patients" population)

| | | 1 1 / | |
|---------|------------|-----------------|-----------------|
| | Proportion | Lower 95% limit | Upper 95% limit |
| CR rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.15 CR rate estimates by the Lugano classification response criteria (Investigator assessment and "Per Protocol Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------|------------|-----------------|-----------------|
| CR rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.16 CR rate estimates by the Lugano classification response criteria (Investigator assessment and "All Evaluable Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------|------------|-----------------|-----------------|
| CR rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.17 CR rate estimates by the Lugano classification response criteria (Investigator assessment and "All Treated Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|---------|------------|-----------------|-----------------|
| CR rate | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.18 Duration of response (Independent Review assessment and "All Responder Patients" population)

| N | X |
|------------|-----|
| Events | X |
| Censored | X |
| Median DoR | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.18)

Table 11.3.2.19 Duration of response (Investigator assessment and "All Responder Patients" population)

| N | X |
|------------|-----|
| Events | X |
| Censored | X |
| Median DoR | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.19)

Table 11.3.2.20 Time to response (Independent Review assessment and "All Responder Patients" population)

| 1 delication propriated ( | |
|---------------------------|-----|
| N | X |
| Median | X |
| Minimum | X |
| Maximum | X.X |

Table 11.3.2.21 Time to response (Investigator assessment and "All Responder Patients" population)

| N | X |
|---------|-----|
| Median | X |
| Minimum | X |
| Maximum | X.X |

Table 11.3.2.22 PFS (Independent Review assessment and "Per Protocol Patients" population)

| N | X |
|------------------|-----|
| Events | X |
| Censored | X |
| Median PFS | X.X |
| PFS at 6 months | X.X |
| PFS at 12 months | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.22)

Table 11.3.2.23 PFS (Independent Review assessment and "All Evaluable Patients" population)

| N | X |
|------------------|-----|
| Events | X |
| Censored | X |
| Median PFS | X.X |
| PFS at 6 months | X.X |
| PFS at 12 months | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.23)

Table 11.3.2.24 PFS (Independent Review assessment and "All Treated Patients" population)

| N | X |
|------------------|-----|
| Events | X |
| Censored | X |
| Median PFS | X.X |
| PFS at 6 months | X.X |
| PFS at 12 months | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.24)

Table 11.3.2.25 PFS (Investigator assessment and "Per Protocol Patients" population)

| N | X |
|------------------|-----|
| Events | X |
| Censored | X |
| Median PFS | X.X |
| PFS at 6 months | X.X |
| PFS at 12 months | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.25)

Table 11.3.2.26 PFS (Investigator assessment and "All Evaluable Patients" population)

| N | X |
|------------------|-----|
| Events | X |
| Censored | X |
| Median PFS | X.X |
| PFS at 6 months | X.X |
| PFS at 12 months | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.26)

Table 11.3.2.27 PFS (Investigator assessment and "All Treated Patients" population)

| N | X |
|------------------|-----|
| Events | X |
| Censored | X |
| Median PFS | X.X |
| PFS at 6 months | X.X |
| PFS at 12 months | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.27)

Table 11.3.2.28 PFS – Concordance between Independent Review assessment and Investigator assessment ("Per Protocol Patients" population)

| investigator assessment ( Tel Trotocol Latients population) | | |
|-------------------------------------------------------------|---|---|
| | N | % |
| Event by investigator | | |
| Agreement on event | | |
| Same date | | |
| Later date | | |
| Earlier date | | |
| Censored by investigator | | |
| Agreement on censoring | | |
| Same date | | |
| Different date | | |
| Agreement on status | | |
| Agreement on status and date | | |

Table 11.3.2.29 Intra-patient PFS/TTP ratio (Independent Review assessment and "Per Protocol Patients" population)

| Ratio | | |
|----------------|---|-----|
| | N | % |
| ≤1.33<br>>1.22 | X | X.X |
| >1.33 | | |

Table 11.3.2.30 Intra-patient PFS/TTP ratio (Independent Review assessment and "All Evaluable Patients" population)

| | , | | |
|-------|---|---|-----|
| Ratio | | | |
| | | N | % |
| ≤1.33 | | X | X.X |
| >1.33 | | | |

Table 11.3.2.31 Intra-patient PFS/TTP ratio (Independent Review assessment and "All Treated Patients" population)

| Ratio | | |
|----------------|---|-----|
| | N | % |
| ≤1.33<br>>1.22 | X | X.X |
| >1.33 | | |

Table 11.3.2.32 Intra-patient PFS/TTP ratio estimates (Independent Review assessment and "Per Protocol Patients" population)

| | 1 1 / | | |
|-------|------------|-----------------|-----------------|
| | Proportion | Lower 95% limit | Upper 95% limit |
| Ratio | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval
Table 11.3.2.33 Intra-patient PFS/TTP ratio estimates (Independent Review assessment and "All Evaluable Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|-------|------------|-----------------|-----------------|
| Ratio | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

# Table 11.3.2.34 Intra-patient PFS/TTP ratio estimates (Independent Review assessment and "All Treated Patients" population)

| 1 | 1 / | | |
|-------|------------|-----------------|-----------------|
| | Proportion | Lower 95% limit | Upper 95% limit |
| Ratio | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

Table 11.3.2.35 Intra-patient PFS/TTP ratio (Investigator assessment and "Per Protocol Patients" population)

| Ratio | | |
|-------|---|-----|
| | N | % |
| ≤1.33 | X | X.X |
| >1.33 | | |

# Table 11.3.2.36 Intra-patient PFS/TTP ratio (Investigator assessment and "All Evaluable Patients" population)

| Ratio | | |
|----------------|---|-----|
| | N | % |
| ≤1.33<br>>1.22 | X | X.X |
| >1.33 | ļ | |

# Table 11.3.2.37 Intra-patient PFS/TTP ratio (Investigator assessment and "All Treated Patients" population)

| Ratio | | |
|-------|---|-----|
| | N | % |
| ≤1.33 | X | X.X |
| >1.33 | | |

# Table 11.3.2.38 Intra-patient PFS/TTP ratio estimates (Investigator assessment and "Per Protocol Patients" population)

| | D (: | Lawar 050/ limit | Umper 050/ limit |
|-------|------------|------------------|------------------|
| | Proportion | Lower 95% limit | Upper 95% limit |
| Ratio | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

# Table 11.3.2.39 Intra-patient PFS/TTP ratio estimates (Investigator assessment and "All Evaluable Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|-------|------------|-----------------|-----------------|
| Ratio | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

# Table 11.3.2.40 Intra-patient PFS/TTP ratio estimates (Investigator assessment and "All Treated Patients" population)

| | Proportion | Lower 95% limit | Upper 95% limit |
|-------|------------|-----------------|-----------------|
| Ratio | X.X | X.X | X.X |

Binomial exact estimator and 95% confidence interval

## Table 11.3.2.41 OS ("Per Protocol Patients" population)

| N | X |
|-----------------|-----|
| Events | X |
| Censored | X |
| Median OS | X.X |
| OS at 6 months | X.X |
| OS at 12 months | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.41).

## Table 11.3.2.42 OS ("All Evaluable Patients" population)

| N | X |
|-----------------|-----|
| Events | X |
| Censored | X |
| Median OS | X.X |
| OS at 6 months | X.X |
| OS at 12 months | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.42).

## Table 11.3.2.43 OS ("All Treated Patients" population)

| N | X |
|-----------------|-----|
| Events | X |
| Censored | X |
| Median OS | X.X |
| OS at 6 months | X.X |
| OS at 12 months | X.X |

Kaplan-Meier plot will be also shown (Figure 11.3.2.43).

## 11.3.3 Follow-up

Median follow-up assessments will be calculated using the Kaplan-Meier method reversing the censoring values (2). In addition, descriptive median and range will be calculated.

## Table 11.3.3.1 Median FU for PFS

| | Median | 95% CI |
|-----------|--------|---------|
| Follow-up | X.X | X.X-X.X |

Table 11.3.3.2 Descriptive median FU for PFS

| _ | Median | Min | Max |
|-----------|--------|-----|-----|
| Follow-up | X.X | X.X | X.X |

## Table 11.3.3.3 Median FU for OS

| | Median | 95% CI |
|-----------|--------|---------|
| Follow-up | X.X | X.X-X.X |

Table 11.3.3.4 Descriptive median FU for OS

| | Median | Min | Max |
|-----------|--------|-----|-----|
| Follow-up | X.X | X.X | X.X |

## 11.3.4 Multivariate analyses

Table 11.3.4.1 Multivariate analysis of PFS (Independent Review assessment and "Per Protocol Patients" population)

| Analysis of Maximum Likelihood Estimates | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |
| variable Eaber | varaes | D1 | Estimate | Liioi | Square | 11 cmsq | Ratio | Emmes |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.2 Multivariate analysis of PFS (Investigator assessment and "Per Protocol Patients" population)

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.3 Multivariate analysis of PFS (Independent Review assessment and "All Evaluable Patients" population)

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.4 Multivariate analysis of PFS (Investigator assessment and "All EvaluablePatients" population)

| E + WI WWO I GI W | riving pop | 0,10,00 | 011) | | | | | |
|---|---|---|---|---|---|---|---|---|
| Analysis of Maximum Likelihood Estimates | | | | | | | | |
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.5 Multivariate analysis of PFS (Independent Review assessment and "All Treated Patients" population)

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Hazard<br>Ratio | 95% Hazard<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.6 Multivariate analysis of PFS (Investigator assessment and "All Treated Patients" population)

| | Analysis of Maximum Likalihood Estimates | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Analysis of Maximum Likelihood Estimates | | | | | | | | |
| | | | | | | | | | 95% Hazard<br>Ratio |
| | | Variable | | Parameter | Standard | Chi- | | Hazard | Confidence |
| Var | riable Label | values | DF | Estimate | Error | Square | Pr > ChiSq | Ratio | Limits |
| | | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.7 Multivariate analysis of ORR (Independent Review assessment and "Per Protocol Patients" population)

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.8 Multivariate analysis of ORR (Investigator assessment and "Per Protocol Patients" population)

| Tatients po | Julation | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Analysis of Maximum Likelihood Estimates | | | | | | | | |
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.9 Multivariate analysis of ORR (Independent Review assessment and "All Evaluable Patients" population)

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | Analysis of M | laximum Like | elihood Esti | mates | | |
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.10 Multivariate analysis of ORR (Investigator assessment and "All Evaluable Patients" population)

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.11 Multivariate analysis of ORR (Independent Review assessment and "All Treated Patients" population)

| Analysis of Maximum Likelihood Estimates | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.12 Multivariate analysis of ORR (Investigator assessment and "All Treated Patients" population)

| Tatients pol | Julution | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Analysis of Maximum Likelihood Estimates | | | | | | | |
| Variable Label | Variable values | DF | Parameter<br>Estimate | Standard<br>Error | Chi-<br>Square | Pr > ChiSq | Odds<br>Ratio | 95% Odds<br>Ratio<br>Confidence<br>Limits |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11 3 4 13 Multivariate analysis of OS ("Per Protocol Patients" population)

| 14010 11.5. | Table 11.5.4.15 With variate analysis of OS (1 of 1 follocoff attents population) | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Analysis of Maximum Likelihood Estimates | | | | | | | |
| Variable Label | Variable values | DF | Parameter<br>Estimate | | _ | Pr > ChiSq | Hazard<br>Ratio | |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.14 Multivariate analysis of OS ("All Evaluable Patients" population)

| | Analysis of Maximum Likelihood Estimates | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable I | Label | Variable<br>values | DF | Parameter<br>Estimate | | _ | Pr > ChiSq | Hazard<br>Ratio | |
| | | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

Table 11.3.4.15 Multivariate analysis of OS ("All Treated Patients" population)

| | Analysis of Maximum Likelihood Estimates | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Variable Lab | Variable el values | DF | Parameter<br>Estimate | | | Pr > ChiSq | Hazard<br>Ratio | |
| | | | X.X | X.X | X.X | X.XXXX | X.X | X.X-X.X |

List of covariates in section 6.2.2

## 11.3.5 Best reduction in sum of the product of the diameters lesions

Table 11.3.5.1 Best reduction in sum of product of diameters from baseline

| SPD | N | Median | Mean | StD | Min | Max |
|-----|---|--------|------|-----|-----|-----|
| | X | X.X | X.X | X.X | X.X | X.X |

Waterfall plot (Figure 11.3.5.1) will be also shown for all patients with at one disease assessment after treatment.

## 11.3.6 Characteristics of responders

A summary of the main characteristics of patients showing clinical benefit, defined as patients with PR or better as best response or SD longer than 6 months assessed by Independent Review or by Investigators will be shown.

Listing 11.3.6.1 Characteristics of patients with clinical benefit.

| | | | , | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient id. | Gender<br>PS<br>Age | Ann-<br>Arbor<br>stage | Bulky<br>Lesion | Relapsed /<br>Refractory | IPI | PAI | PIAI | No.<br>of<br>prior<br>lines | Cycles received | Best<br>response<br>Lugano<br>(IA) | Best<br>response<br>Lugano<br>(IR) | Best<br>PET<br>SUV<br>reduction<br>(%) | PFS<br>(IA) | DR<br>(IA) | PFS<br>(IR) | DR<br>(IR) | os |

IR- Independent review IA- Investigator assessment

# 12 Safety Analysis

Safety analysis will be carried out on the "All Treated Patients" population.

## 12.1 Extent of exposure

## 12.1.1 Treatment administration

Table 12.1.1.1 Number of cycles administered and dose intensity

| No. of cycles administered per patient | N | % |
|-----------------------------------------|-----|-------|
| 1 | X | X.X |
| 2 | | |
| 3 | | |
| ••• | | |
| Median (range) | X.X | (X-X) |
| Time on treatment (weeks) | | |
| Median | X | ī.X |
| Range | X.X | -X.X |
| Plitidepsin cumulative dose (mg/m²) | | |
| Median | X | i.X |
| Range | X.X | -X.X |
| Plitidepsin dose intensity (mg/m²/wk) | | |
| Median | X | X |
| Range | X.X | -X.X |
| Plitidepsin relative dose intensity (%) | | |
| Median | X.X | |
| Range | X.X | -X.X |

## 12.1.2 Cycle delays

## 12.1.2.1 Number of patients and cycles with dosing delay, any relationship

Listing 12.1.2.1.1 Delays

| Patient id. | Cycle | Day | Previous cycle | Previous cycle start date | Delayed cycle | Delayed<br>cycle start<br>date | Dose Delay calculated. (days) | Reason<br>for dose<br>delay | Dose<br>Delay<br>Spec. |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | X | | |

Table 12.1.2.1.2 Number of patients and cycles with dosing delay, any relationship

| | N | % |
|-----------------------------------------------------|---|-----|
| No. of patients treated | X | X.X |
| No. of patients susceptible to have a dosing delay* | | |
| No. of patients with any dose delay** | | |
| No. of cycles administered | | |
| No. of cycles susceptible to be delayed*** | | |
| No. of cycles with dosing delay**** | | |
| No. of patients with | | |
| No cycles delayed | | |
| 1 cycle delayed | | |
| 2 cycles delayed | | |
| ≥ 3 cycles delayed | | |

<sup>(\*)</sup> All patients with more than one cycle. (\*\*) Denominator = Number of patients susceptible to have a dosing delay (\*\*\*) All cycles excluding first cycle. (\*\*\*\*) Denominator = Number of cycles susceptible to be delayed

Table 12.1.2.1.3 Number of patients and cycles with dosing delay according to the relationship

| | Treatm | ent-related | Non-treatment-related | |
|---|---|---|---|---|
| | N | % | N | % |
| No. of patients with * 1 cycle delayed 2 cycles delayed ≥ 3 cycles delayed | X | X.X | | |
| No. of cycles with dosing delay** | | | | |

<sup>(\*)</sup> Denominator = Number of patients susceptible to have a dosing delay (\*\*) Denominator= Number of cycles susceptible to be delayed.

Table 12.1.2.1.4 Length of dosing delay.

| | Treatment-related | | Non-treatn | Total | | |
|---|---|---|---|---|---|---|
| Length of delay Median (range) | | | | | | |
| Length of delay | N | % | N | % | N | % |
| <= 7 days | X | X.X | | | | |
| >7 days and <=14 days | | | | | | |
| > 14 days | | | | | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to be delayed.

Listing 12.1.2.1.5 Cycle delays due to AEs

| Patient id. | Cycle | Delay<br>reason<br>according<br>to Exposure<br>form | Preferred term code | Adverse<br>event<br>reported<br>(verbatim) | Grade | Relationship | Onset date | Resolved date | Significant consequences |
|---|---|---|---|---|---|---|---|---|---|

AEs with action = 'Dose delayed' or 'Reduced and delayed'.

### 12.1.3 Dose omissions

Listing 12.1.3.1 Dose omissions

| Patient id. | Cycle | Day | Cycle start date | Reason for dose omission | Dose omission Spec. |
|---|---|---|---|---|---|

Table 12.1.3.2 Number of patients and cycles with dose omitted, any relationship

| | N | % |
|-------------------------------------------------------------------|---|-----|
| No. of patients treated | X | X.X |
| No. of patients susceptible to have a dose omission * | | |
| No. of patients with any dose omitted ** | | |
| No. of patients with **: | | |
| No plitidepsin omissions | | |
| 1 cycle with plitidepsin dose omitted | | |
| 2 cycles with plitidepsin dose omitted | | |
| ≥ 3 cycles with plitidepsin dose omitted | | |
| No. of cycles administered | | |
| No. of cycles susceptible to have any dose omitted*** | | |
| No. of cycles with plitidepsin dosing omitted**** | | |
| No. of cycles with plitidepsin dosing omitted (treatment-related) | | |

<sup>(\*)</sup> All patients with more than one infusion. (\*\*) Denominator = Number of patients susceptible to have a dose omission (\*\*\*) All cycles excluding first cycle. (\*\*\*\*) Denominator = Number of cycles susceptible to have a dose omission NA: Not applicable

Table 12.1.3.3 Number of cycles with treatment-related dose omission by patient

| | N | % |
|------------------------------------------------------------|---|-----|
| No. of patients with: | X | X.X |
| No omission | | |
| 1 cycle with treatment-related plitidepsin dose omitted | | |
| 2 cycles with treatment-related plitidepsin dose omitted | | |
| ≥ 3 cycles with treatment-related plitidepsin dose omitted | | |

Denominator= Number of patients that were on treatment on day 8 of cycle 1.

NA: Not applicable

## Table 12.1.3.4 Reasons for dose omissions

| Reasons for omissions | N | % |
|-----------------------|---|-----|
| Treatment-related | X | X.X |
| Non-treatment-related | | |

NA: Not applicable

Listing 12.1.3.5 Dose omissions due to AEs

| Patient id. | Cycle | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset<br>date | Resolved<br>date | Significant consequences |
|---|---|---|---|---|---|---|---|---|

AEs with action = 'Dose skipped" on day 8 or 15.

#### 12.1.4 Dose reductions

All dose reductions should be considered and described, specifying the reason for reduction (drug related, non-drug related or other causes).

Listing 12.1.4.1 Dose reductions

| Patient id. | Cycle | Day | Cycle start date | Previous dose | Reduced dose | Reason for dose reduction | Dose reduction Spec. |
|---|---|---|---|---|---|---|---|

Table 12.1.4.2 Number of patients and cycles with dose reduction, any relationship

| | N | % |
|-----------------------------------------------------------------|---|-----|
| No. of patients treated | X | X.X |
| No. of patients susceptible to have a dose reduced* | | |
| No. of patients with any dose reduced** | | |
| No. of patients with**: | | |
| No plitidepsin reduction | | |
| 1 cycle with plitidepsin dose reduced | | |
| 2 cycles with plitidepsin dose reduced | | |
| No. of cycles administered | | |
| No. of cycles susceptible to have any dose reduced*** | | |
| No. of cycles with plitidepsin dose reduced **** | | |
| No. of cycles with plitidepsin dose reduced (Treatment-related) | | |

(\*) All patients with more than one infusion. (\*\*) Denominator = Number of patients susceptible to have a dose reduced (\*\*\*) All cycles excluding first cycle of those patients who have only received the first infusion. (\*\*\*\*) Denominator= Number of cycles susceptible to have a dose omission

NA: Not applicable

Table 12.1.4.3 Number of patients and cycles with dose reduction according to the relationship

| relationship | | |
|-------------------------------------|---|-----|
| Reasons for reductions | N | % |
| No. of cycles with dose reductions* | | |
| Treatment-related | X | X.X |
| Non-treatment-related | | |

<sup>(\*)</sup> Denominator= Number of cycles susceptible to have a dose omission

NA: Not applicable

Listing 12.1.4.4 Dose reductions due to AEs

| Patient id. | Cycle | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset date | Resolved date | Significant consequences |
|---|---|---|---|---|---|---|---|---|

AEs with action = 'Dose reduced/adjusted' or 'Reduced and delayed'.

## 12.1.5 Infusions temporarily interrupted

A listing of the patients who had infusions temporarily interrupted with the corresponding reasons will be provided.

Listing 12.1.5.1 Interrupted Infusions listing.

| Patient id. | Cycle | Infusion | Interrupted | Reason |
|-------------|-------|----------|-------------|--------|
| | | | Yes | |

## 12.1.6 Prophylactic medication administration

A listing of the patients who have not received Ondansetron, Diphenhydramine and Ranitidine or equivalents with the corresponding reasons will be reported.

Listing 12.1.6.1 Patients and cycles without prophylactic medication administration

| Patient id. | Cycle | Infusion | Prophylactic medication not taken* | Reason |
|-------------|-------|----------|------------------------------------|--------|

<sup>(\*)</sup> Ondansetron, diphenhydramine or ranitidine.

# 12.2 Adverse Events (AEs)

# 12.2.1 Display of adverse events

Table 12.2.1.1 Summary of adverse events.

| | N (%) |
|------------------------------------------------------------|---------|
| Patients with at least one AE regardless relationship | X (X.X) |
| Any treatment-related AE | |
| Any grade 3/4 AE | |
| Any grade 3/4 treatment-related AE | |
| Any SAE in DB | |
| Any treatment-related SAE | |
| Any grade 3/4 SAE | |
| Any grade 3/4 treatment-related SAE | |
| AEs leading to death | |
| AEs treatment-related leading to death | |
| AEs leading to dose delay | |
| AEs leading to dose reduction | |
| AEs leading to treatment discontinuation | |
| AEs treatment-related leading to treatment discontinuation | |

Table 12.2.1.2 Evolution of lymphoma-related AEs at baseline

| | | <u> </u> | | Worst grade per patient | | | | | - | Гotal |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | 0 | | 1 | | | | Total |
| | | | N | % | N | % | N | % | N | % |
| | Fatigue | Grade 0 | X | X.X | X | X.X | X | X.X | X | X.X |
| Bone Pain Bone Pain | Grade 1 | | | | | | | | | |
| | Grade 0 | | | | | | | | | |
| | Grade 1 | | | | | | | | | |
| sase | | | | | | | | | | |
| Щ | Myopathy | Grade 0 | | | | | | | | |
| | Grade 1 | | | | | | | | | |
| | | <u> </u> | | | | | | | | |

Table 12.2.1.3 Treatment-related\* adverse events. Worst grade by patient

| | | Gr | ade<br>1 | <br>Gr | ade<br>4 | Al | 1** |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic | Anemia NOS | X | X.X | X | X.X | X | X.X |
| system disorders | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> or Uknown relationship (\*\*) Any grade

Table 12.2.1.4 Treatment-related\* adverse events. Worst grade by cycle

| | | Grade | | Grade<br>4 | | All** | | |
|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | | N | % | N | % |
| Blood and lymphatic | Anemia NOS | X | X.X | | X | X.X | X | X.X |
| system disorders | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | |

<sup>(\*)</sup> or Uknown relationship (\*\*) Any grade

Table 12.2.1.5 Adverse Events regardless of relationship. Worst grade by patient

| Twell 12:2:1:0 114 + 0150 2 + 0116 10 Millions of 1010010 mpt. ++ 0150 Brown of position | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Grade<br>1 | | Grade Grade 4 | | ade<br>4 | All* | |
| SOC | Preferred Term | N | % | | N | % | N | % |
| Blood and lymphatic | Anemia NOS | X | X.X | | X | X.X | X | X.X |
| system disorders | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.2.1.6 Adverse Events regardless of relationship. Worst grade by cycle

| | | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic | Anemia NOS | X | X.X | X | X.X | X | X.X |
| system disorders | ••• | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.2.1.7 Treatment-related\* grade 3-4 adverse events. Worst grade by patient

| Patient id. | SOC Name | Preferred term | Grade |
|-------------|----------|----------------|-------|

<sup>(\*)</sup> or Uknown relationship

Listing 12.2.1.8 Treatment-related\* grade 3-4 adverse events. Worst grade by cycle

| | <u> </u> | | · · J · · J · · | | |
|-------------|----------|-------|-----------------|----------------|-------|
| Patient id. | | Cycle | SOC Name | Preferred term | Grade |

<sup>(\*)</sup> or Uknown relationship

Listing 12.2.1.9 Adverse Events grade 3-4 regardless of relationship. Worst grade by patient

| Patient id. | SOC Name | Preferred term | Grade |
|-------------|----------|----------------|-------|

Listing 12.2.1.10 Adverse Events grade 3-4 regardless of relationship. Worst grade by cycle

| | - · · · · · · | | , | | |
|-------------|---------------|-------|----------|----------------|-------|
| Patient id. | | Cycle | SOC Name | Preferred term | Grade |

At the time of the analysis, if appropriate, grouping of similar or clinically related items will be made.

### 12.3 Serious Adverse Events and deaths.

### 12.3.1 Serious Adverse Events

Table 12.3.1.1 Treatment-related\* SAEs. Worst grade by patient

| | | Gr | ade<br>1 | <br>Gr | ade<br>4 | Al | 1** |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic | Anemia NOS | X | X.X | X | X.X | X | X.X |
| system disorders | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | |

<sup>(\*)</sup> or Uknown relationship (\*\*) Any grade

Table 12.3.1.2 Treatment-related\* SAEs. Worst grade by cycle

| | | Gı | rade<br>1 | ••• | Gr | ade<br>4 | Al | 1** |
|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | | N | % | N | % |
| Blood and lymphatic | Anemia NOS | X | X.X | | X | X.X | X | X.X |
| system disorders | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | |

<sup>(\*)</sup> or Uknown relationship (\*\*) Any grade

Table 12.3.1.3 SAEs regardless of relationship. Worst grade by patient

| | | - | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | | N | % | <br>N | % | N | % |
| Blood and lymphatic | Anemia NOS | | X | X.X | X | X.X | X | X.X |
| system disorders | | | | | | | | |
| Cardiac disorders | Arrhythmia NOS | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.3.1.4 SAEs regardless of relationship. Worst grade by cycle

| | | Gr | ade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|---|---|---|---|---|---|---|---|
| SOC | Preferred Term | N | % | <br>N | % | N | % |
| Blood and lymphatic system disorders | Anemia NOS | X | X.X | X | X.X | X | X.X |
| Cardiac disorders | Arrhythmia NOS | | | | | | |
| (d) 1 | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.3.1.5 SAEs

| | , | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Patient id. | Cycle | Preferred term code | Adverse<br>event<br>reported<br>(verbatim) | Status | Grade | Relationship | Onset date | Resolved<br>date | Action | Serious Criteria |

SAEs narratives will be provided by the pharmacovigilance department.

#### 12.3.2 Deaths

Table 12.3.2.1 Cause of death

| Reason* | N | % |
|---------------------------------|---|-----|
| Malignant disease | X | X.X |
| Treatment-related adverse event | | |
| Other | | |
| Total | | |

<sup>(\*)</sup> Denominator=Number of patients who died

Listing 12.3.2.2 Deaths

| Patient id. | Death date | Cause | Comments | Autopsy | Autopsy report<br>available | Number of cycles administered | Last infusion date | Time on treatment* | Time from<br>Last dose** |
|---|---|---|---|---|---|---|---|---|---|

<sup>(\*)</sup>Time on treatment: defined as last infusion date plus 30 days, or date of death or subsequent therapy (whichever comes first) minus first infusion date. (\*\*)Time from last dose defined as death date minus last infusion date.

Listing 12.3.2.3 Deaths due to AEs

| Patient id. | Cycle | Preferred term code | Adverse event reported (verbatim) | Grade | Relationship | Onset<br>date | Resolved date | Action |
|---|---|---|---|---|---|---|---|---|

### 12.4 Clinical laboratory evaluation

## 12.4.1 Hematological abnormalities

Hematological toxicities classified according to the NCI-CTCAE will be calculated for all cycles. The worst grade reached by each patient during treatment will be also calculated.

If serious toxicities happen, special follow-up, with descriptives and graphs (boxplots, line plots) will be made to find out the pattern of thrombocytopenia and neutropenia within and between the different cycles.

Table 12.4.1.1 Hematological abnormalities during treatment, worst grade per patient

| | N | Grade<br>1 | | | Grade<br>4 | | All* | |
|---|---|---|---|---|---|---|---|---|
| | N | N | % | ••• | N | % | N | % |
| Leukopenia | X | X | X.X | | X | X.X | X | X.X |
| Anemia | | | | | | | | |
| Thrombocytopenia | | | | | | | | |
| Neutropenia | | | | | | | | |
| Lymphopenia | | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.4.1.2 Hematological abnormalities during treatment, worst grade per cycle

| | N | N Grade | | ••• | Grade 4 | | All* | |
|------------------|---|---------|-----|-----|---------|-----|------|-----|
| | N | N | % | | N | % | N | % |
| Leukopenia | X | X | X.X | | X | X.X | X | X.X |
| Anemia | | | | | | | | |
| Thrombocytopenia | | | | | | | | |
| Neutropenia | | | | | | | | |
| Lymphopenia | | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.4.1.3 Grade 3-4 hematological abnormalities during treatment. Worst grade per patient

| Patient id. | Test | Grade |
|-------------|------|-------|

Listing 12.4.1.4 Grade 3-4 hematological abnormalities during treatment. Worst grade per cycle

| Patient id. | Test | Grade |
|-------------|------|-------|

Listing 12.4.1.5 Hematological tests not assessed at any treatment visit per patient

| Patient id. | Lab. test |
|-------------|-----------|

Listing 12.4.1.6 Hematological tests not assessed by patient and cycle

| | | <i>J</i> 1 | 2 |
|---------|-----|------------|-----------|
| Patient | id. | Cycle | Lab. test |
| | | _ | |

Table 12.4.1.7 Platelets and RBC transfusions during the study

| | | Platelet | Platelets (Units) | | Cells (Units) |
|---|---|---|---|---|---|
| | | N | (%) | N | (%) |
| | 0 transfusions | X | X.X | X | X.X |
| Platelets (Units) | 1 transfusion | | | | |
| Flatelets (Ollits) | | | | | |
| | Median (range) | | | | |
| | 0 transfusions | | | | |
| Red Blood Cells (Units) | 1 transfusion | | | | |
| | Median (range) | | | | |

These tables will be complemented with plots for the median nadir of neutrophils (Figure 12.4.1.8), platelets count (Figure 12.4.1.9) and hemoglobin values (Figure 12.4.1.10) by cycle along the treatment. Furthermore, if appropriate, graphs of the intercycle time course of neutropenia and thrombocytopenia will be provided. Eventually, graphs comparing the time course during the first and second cycle will be created.

#### 12.4.2 Biochemical abnormalities

Grades of liver toxicity and intercycle pattern of creatinine, CPK, bilirubin, transaminases increase and alkaline phosphatase increase during a cycle will be calculated, as it is explained in the corresponding section for hematological toxicities.

Table 12.4.2.1 Biochemical abnormalities during treatment, worst grade per patient

| | N | | rade<br>1 | | | ade<br>4 | Al | 11* |
|--------------------------|---|---|-----------|-----|---|----------|----|-----|
| | N | N | % | ••• | N | % | N | % |
| AST increase | X | X | X.X | | X | X.X | X | X.X |
| ALT increase | | | | | | | | |
| Total bilirubin increase | | | | | | | | |
| ALP increase | | | | | | | | |
| Creatinine increase | | | | | | | | |
| CPK increase | | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.4.2.2 Biochemical abnormalities during treatment, worst grade per cycle

| | N | G | rade<br>1 | <br>Gr | ade<br>4 | A | 11* |
|--------------------------|---|---|-----------|--------|----------|---|-----|
| | N | N | % | <br>N | % | N | % |
| AST increase | X | X | X.X | X | X.X | X | X.X |
| ALT increase | | | | | | | |
| Total bilirubin increase | | | | | | | |
| ALP increase | | | | | | | |
| Creatinine increase | | | | | | | |
| CPK increase | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.4.2.3 Grade 3-4 biochemical abnormalities during treatment. Worst grade per patient

| P | | |
|-------------|------|-------|
| Patient id. | Test | Grade |

# Listing 12.4.2.4 Grade 3-4 biochemical abnormalities during treatment. Worst grade per cycle

| Patient id. | Cycle | Test | Grade |
|-------------|-------|------|-------|

Listing 12.4.2.5 Biochemical tests not assessed at any treatment visit by patient

| | the state of the s |
|---|---|
| Patient id. | Lab. test |

Listing 12.4.2.6 Biochemical tests not assessed by patient and cycle

| Patient id. | Cycle | Lab. test |
|-------------|-------|-----------|
| | • | |

These tables will be complemented with plots for the median peak of ALT (Figure 12.4.2.7), AST (Figure 12.4.2.8) and CPK values (Figure 12.4.2.9) by cycle along the treatment. If appropriate, graphs of the intercycle time course of ALT, AST and CPK will be provided.

## 12.4.3 Other metabolic parameters

Table 12.4.3.1 Metabolic abnormalities during treatment, worst grade per patient

| | N | Gr | ade<br>1 | <br>Gra | ade<br>1 | Al | 11* |
|-----------------|---|----|----------|---------|----------|----|-----|
| | N | N | % | <br>N | % | N | % |
| Hyperglycemia | X | X | X.X | X | X.X | X | X.X |
| Hypoglycemia | | | | | | | |
| Hypoalbuminemia | | | | | | | |

<sup>(\*)</sup> Any grade

Table 12.4.3.2 Metabolic abnormalities during treatment, worst grade per cycle

| | N | Gr | ade<br>1 | | Gra | ade<br>I | A | 11* |
|-----------------|---|----|----------|-----|-----|----------|---|-----|
| | N | N | % | ••• | N | % | N | % |
| Hyperglycemia | X | X | X.X | | X | X.X | X | X.X |
| Hypoglycemia | | | | | | | | |
| Hypoalbuminemia | | | | | | | | |

<sup>(\*)</sup> Any grade

Listing 12.4.3.3 Grade 3-4 metabolic abnormalities during treatment. Worst grade by patient

| _ r ***** | | |
|-------------|------|-------|
| Patient id. | Test | Grade |

Listing 12.4.3.4 Grade 3-4 metabolic abnormalities during treatment. Worst grade by cycle

| Patient id. | Cycle | Test | Grade |
|-------------|-------|------|-------|

Listing 12.4.3.5 Metabolic tests not assessed at any treatment visit by patient

| Patient id. | Lab. test |
|-------------|-----------|

Listing 12.4.3.6 Metabolic tests not assessed by patient and cycle

| | | - 0 |
|-------------|-------|-----------|
| Patient id. | Cycle | Lab. test |

# 12.4.4 Laboratory values over time

In this section, grades 3-4 hematological and liver enzyme abnormalities will be displayed according to the cycle in which they occurred.

Table 12.4.4.1 Evolution of hematological abnormalities from baseline, worst case per patient.

| | | | Wo | orst grade per pa | tient | Total |
|---|---|---|---|---|---|---|
| | | | 0 | 1 | | Total |
| | Neutropenia | Grade 0 | | | | |
| | | Grade 1 | | | | |
| ine | Thrombocytopenia | Grade 0 | | | | |
| Baseline | | Grade 1 | | | | |
| Ba | | | | | | |
| | | Grade 0 | | | | |
| | | Grade 1 | | | | |

Table 12.4.4.2 Evolution of transaminases abnormalities from BL, worst case per patient.

| | | | | W | orst grade | per pat | ient | | To | to1 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | ( | ) | 1 | | | | 10 | tai |
| | | | N | % | N | % | N | % | N | % |
| | AST increase | X | X.X | X | X.X | | | X | X.X | |
| | | Grade 1 | | | | | | | | |
| ne | ALT increase | Grade 0 | | | | | | | | |
| Baseline | | Grade 1 | | | | | | | | |
| Ba | | | | | | | | | | |
| | | Grade 0 | | | | | | | | |
| | | Grade 1 | | | | | | | | |
| İ | | | | | | | | | | |

Table 12.4.4.3 Grade 3-4 laboratory abnormalities in the first cycle and in all other cycles

| | | | | | <u> </u> | |
|---|---|---|---|---|---|---|
| Laboratory | | Cycle 1 | | Cycle>1 | | |
| abnormalities | No. of cycles evaluated | No. of cycles grade 3-4 | % | No. of cycles evaluated | No. of cycles grade 3-4 | % |
| Thrombocytopenia | X | X | X.X | X | X | X.X |
| Neutropenia | | | | | | |
| ALP | | | | | | |
| Total bilirubin | | | | | | |
| AST | | | | | | |
| ALT | | | | | | |
| СРК | | | | | | |

Table 12.4.4.4 Hemtological time-course pattern

| | Onset<br>day | Days in grade 3- | Day of 1 | recovery to g | grade 2 | Da | ays to recove | ery |
|---|---|---|---|---|---|---|---|---|
| Laboratory abnormalities | grade 3- | 4 | <=28 | 29-35 | >35 | <=28 | 29-35 | >35 |
| Anemia | X (X-X) | X (X-X) | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) |
| Neutropenia | | | | | | | | |
| Thrombocytopenia | | | | | | | | |

Table 12.4.4.5 ALT/AST/CPK time-course pattern

| | Onset<br>day | Days in grade 3- | Day of re | covery to 2.5 | 5 x ULN | Da | ays to recove | ery |
|---|---|---|---|---|---|---|---|---|
| Laboratory abnormalities | grade 3- | 4 | <=28 | 29-35 | >35 | <=28 | 29-35 | >35 |
| ALT | X (X-X) | X (X-X) | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) |
| AST | | | | | | | | |
| СРК | | | | | | | | |

## 12.5 Vital signs, physical findings, LVEF, ECG and other tests related to safety

## 12.5.1 Vital signs and physical findings

Table 12.5.1.1 ECOG performance status during the study

| | | Cycle/PS* | | | |
|-------------|---|-----------|---|---|----|
| | 0 | 1 | 2 | 3 | •• |
| Patient id. | | | | | |

<sup>(\*)</sup> Worst ECOG PS of the cycle determinations.

Table 12.5.1.2 Weight by patient per cycle

| | | Cycle/Weight | | | |
|-------------|-----------|------------------|------|------|----------|
| | 0<br>(kg) | 0 1* 2* 3* | | | |
| Patient id. | (Kg) | (70) | (70) | (70) | <u> </u> |
| | X.X | X.X | X.X | X.X | |

<sup>(\*) %</sup> of changes respect to baseline

## 12.5.2 LVEF, ECG and other related tests

Listing 12.5.2.1 Electrocardiogram results. Evolution during the study.

| Eisting 12.5.2.1 Electrocardiogram results. Evolution during the study. | | |
|---|---|---|
| Patient id. | Cycle | ECG result |

Listing 12.5.2.2 LVEF evolution during the study.

| Patient id. | | LVEF(%) | |
|---------------|--------------|--------------|-------------------|
| i atient id. | Baseline* | Minimun* | End of treatment* |
| | X.X | X.X | X.X |
| Median(Range) | X.X(X.X-X.X) | X.X(X.X-X.X) | X.X(X.X-X.X) |

<sup>(\*)</sup> LVEF (%) value and method

Listing 12.5.2.3 Median change in LVEF.

| Cycles | LVEF |
|------------------|--------------|
| Baseline | X.X(X.X-X.X) |
| Minimun | X.X(X.X-X.X) |
| End of treatment | X.X(X.X-X.X) |

## 12.6 Concomitant therapy / procedures according to the ATC classification.

Table 12.6.1 Concomitant medication during treatment (ATC levels)

| | | 2 | | | |
|---|---|---|---|---|---|
| Medication Term | Medication Term | Medication Term | Preferred Name | | |
| (ATC level 1) | (ATC level 2) | (ATC level 4) | Preferred Name | N | % |
| | | | | X | X.X |

Listing 12.6.2 Patients with EPO or G-CSF.

| Patient id. | Туре | Route | Dose | Unit | Start date | Stop<br>date | Reason | Indication |
|---|---|---|---|---|---|---|---|---|

Listing 12.6.3 Patients with any transfusion during treatment

| Patient | Cycle | Date | Blodd product | Specify | Total units | Irradiated |
|---------|-------|------|---------------|---------|-------------|------------|

Taken from concomitant therapy dataset.

Table 12.6.4 G-CSF, transfusions or EPO during treatment

| | N | % |
|-------------------------------|---|-----|
| G-CSF | X | X.X |
| Platelets transfusions | | |
| Packed red cells transfusions | | |
| Plasma transfusions | | |
| Cryoprecipitates | | |
| Clotting factors | | |
| EPO | | |

Table 12.6.5 Subsequent therapy

| | N | % |
|--------------------------------------|---|-----|
| Type | X | X.X |
| Chemotherapy | | |
| Subsequent chemotherapy agents (ATC) | | |

Table 12.6.6 Time to subsequent therapy or death

| | Arm A | Arm B | Parameter | p-value |
|-------------------------------|-------|-------|--------------|---------|
| N | | | | |
| Events | | | | |
| Censored | | | | |
| Time to subsequent therapy or | | | Log-Rank: | LR: |
| death | | | HR (95% CI): | HR: |

Kaplan-Meier plot will be also shown (Figure 12.6.7)

## 12.7 Safety analysis in special subgroups.

Table 12.7.1 Worst grade 3-4 by patient in special subgroups (Gender)

| | | Male | | | Female | |
|------------------|---|-----------|-----|---|-----------|-----|
| | N | Grade 3-4 | % | N | Grade 3-4 | % |
| Thrombocytopenia | X | X | X.X | X | X | X.X |
| Neutropenia | | | | | | |
| ALP | | | | | | |
| Total bilirubin | | | | | | |
| AST | | | | | | |
| ALT | | | | | | |
| СРК | | | | | | |
| Nausea | | | | | | |
| Vomiting | | | | | | |
| Fatigue | | | | | | |
| Other* | | | | | | |

<sup>(\*)</sup> Any treatment-related toxicity present in >=5% of patients in any group

Table 12.7.2 Worst grade 3-4 by patient in special subgroups (Race)

| | 7 1 | White | <u> </u> | Other | | |
|---|---|---|---|---|---|---|
| | N | Grade 3-4 | % | N | Grade 3-4 | % |
| Thrombocytopenia | X | X | X.X | X | X | X.X |
| Neutropenia | | | | | | |
| ALP | | | | | | |
| Total bilirubin | | | | | | |
| AST | | | | | | |
| ALT | | | | | | |
| СРК | | | | | | |
| Nausea | | | | | | |
| Vomiting | | | | | | |
| Fatigue | | | | | | |
| Other* | | | | | | |
| | y progent in >-50/ | of nationts in any | aroun | | | |

<sup>(\*)</sup>Any treatment-related toxicity present in >=5% of patients in any group

Table 12.7.3 Worst grade 3-4 by patient in special subgroups (Age)

| | <65 years old | | | ≥65 years old | | |
|---|---|---|---|---|---|---|
| | N | Grade 3-4 | % | N | Grade 3-4 | % |
| Thrombocytopenia | X | X | X.X | X | X | X.X |
| Neutropenia | | | | | | |
| ALP | | | | | | |
| Total bilirubin | | | | | | |
| AST | | | | | | |
| ALT | | | | | | |
| СРК | | | | | | |
| Nausea | | | | | | |
| Vomiting | | | | | | |
| Fatigue | | | | | | |
| Other* | | | | | | |

<sup>(\*)</sup>Any treatment-related toxicity present in >=5% of patients in any group

Table 12.7.4 Worst grade 3-4 by patient in special subgroups (BMI)

| | | <30 | | | ≥30 | |
|------------------|---|-----------|-----|---|-----------|-----|
| | N | Grade 3-4 | % | N | Grade 3-4 | % |
| Thrombocytopenia | X | X | X.X | X | X | X.X |
| Neutropenia | | | | | | |
| ALP | | | | | | |
| Total bilirubin | | | | | | |
| AST | | | | | | |
| ALT | | | | | | |
| СРК | | | | | | |
| Nausea | | | | | | |
| Vomiting | | | | | | |
| Fatigue | | | | | | |
| Other* | | | | | | |

<sup>(\*)</sup>Any treatment-related toxicity present in >=5% of patients in any group

#### APPENDIX II

## 13 DB Listings

-Listing 13.1.40: Off study

### CRF Listings.

-Listing 13.1.1: Screening -Listing 13.1.2: Demography -Listing 13.1.3: Contraception and pregnancy test -Listing 13.1.4: Medical history -Listing 13.1.5: Lymphoma history -Listing 13.1.6: Prior radiotherapy -Listing 13.1.7: Prior surgery -Listing 13.1.8: Prior anticancer therapy -Listing 13.1.9: Prophylactic medication -Listing 13.1.10: Drug administration -Listing 13.1.11: Hematology laboratory values -Listing 13.1.12: Coagulation laboratory values -Listing 13.1.13: Biochemical laboratory values -Listing 13.1.14: Other metabolic laboratory values -Listing 13.1.15: Urinary dipstick -Listing 13.1.16: Viral serology -Listing 13.1.17: Coombs Test -Listing 13.1.18: Protein measurements -Listing 13.1.19: Physical examination -Listing 13.1.20: Performance status -Listing 13.1.21: Neurological examination -Listing 13.1.22: Vital signs -Listing 13.1.23: Electrocardiogram -Listing 13.1.24: LVEF -Listing 13.1.25: Bone marrow assessment -Listing 13.1.26: Blood product use -Listing 13.1.27: Adverse events (including signs and symptoms) -Listing 13.1.28: Concomitant medications -Listing 13.1.29: Concomitant procedures -Listing 13.1.30: Other tests/procedures -Listing 13.1.31: Tumor evaluation -Listing 13.1.32: Overall response assessment by cycle -Listing 13.1.33: Best overall response -Listing 13.1.34: End of treatment -Listing 13.1.35: Follow up -Listing 13.1.36: Medical treatment (after end of treatment) -Listing 13.1.37: Surgery procedures (after end of treatment) -Listing 13.1.38: Radiotherapy (after end of treatment) -Listing 13.1.39: Death report form

### APPENDIX II

# 14 Section 16.2 ICH Listings

- -ICH Listing 16.2.1: Discontinued patients
- -ICH Listing 16.2.2: Protocol deviations
- -ICH Listing 16.2.3: Patients excluded from the efficacy analysis
- -ICH Listing 16.2.4: Demographic data
- -ICH Listing 16.2.5: Compliance and-or Drug Concentration Data
- -ICH Listing 16.2.6: Individual Efficacy Response data
- -ICH Listing 16.2.7: Adverse Events
- -ICH Listing 16.2.8: Individual laboratory measurements

# 15 References

- 1. SAS OnlineDoc, V9.
- 2. Parmar M. Machin D. Survival analysis. A practical approach. Wiley, Chichester, 1995.